CLINICAL TRIAL: NCT00383188
Title: A 12-WEEK, PHASE 2A, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO INVESTIGATE THE SAFETY, PHARMACOKINETICS, AND EFFICACY OF PH 797804, ADMINISTERED ORALLY ONCE DAILY IN SUBJECTS WITH ACTIVE RHEUMATOID ARTHRITIS
Brief Title: An Oral p38 Inhibitor Investigating Safety, Efficacy, And PK In Subjects With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A6631007; 2006-003577-27 (EudraCT Number); RA POC (Other: Alias Study Number)
Record Dates: First submitted 2006-09-28; First posted 2006-10-02 (Estimated); Results first posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-07

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis; Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — PH 797804

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Experimental)
  Interventions: Drug: PH-797804
- 3 (Experimental)
  Interventions: Drug: PH-797804
- 4 (Experimental)
  Interventions: Drug: PH-797804
- 5 (Experimental)
  Interventions: Drug: PH-797804

INTERVENTIONS:
Drug: placebo — Capsule, once daily (QD) for 12 weeks
  Arms: 1
Drug: PH-797804 — Capsule, 0.5 mg of PH-797804, once daily (QD) for 12 weeks
  Arms: 2
Drug: PH-797804 — Capsule, 3 mg of PH-797804, once daily (QD) for 12 weeks
  Arms: 3
Drug: PH-797804 — Capsule, 6 mg of PH-797804, once daily (QD) for 12 weeks
  Arms: 4
Drug: PH-797804 — Capsule, 10 mg of PH-797804, once daily (QD) for 12 weeks
  Arms: 5

SUMMARY:
Investigating the safety and tolerability of a p38 inhibitor as monotherapy in subjects who have failed at least 1 DMARD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RA and has failed at least 1 DMARD therapy

Exclusion Criteria:

* Any other inflammatory arthritis and any significant history of acute or chronic infection with immunomodulatory etiology.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2006-12-15 (Actual); Primary Completion 2008-07-01 (Actual); Study Completion 2008-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (48):
- Emeritus Research, Malvern East, Victoria, Australia
- Brazil (4):
  - Centro de Estudos em Terapias Inovadoras, Curitiba, Paraná
  - Hospital de Clínicas da UFPR, Curitiba, Paraná
  - Escola Paulista de Medicina - EPM, São Paulo, São Paulo
  - Hospital Heliópolis - PAM, São Paulo, São Paulo
- Chile (5):
  - Hospital Gustavo Fricke, Viña del Mar, Región de Valparaíso
  - Hospital Regional de Rancagua, Rancagua, Región del Libertador General Bernardo O’Higgins
  - Hospital del Salvador, Santiago, RM
  - Office of Dr. Pedro Miranda, Santiago, RM
  - Hospital Clínica San Borja Arriarán, Santiago, RM
- Czechia (6):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - NZZ Bormed, s.r.o., Ostrava - Trebovice
  - Revmatologicky ustav, Prague
  - Fakultni Thomayerova nemocnice s poliklinikou, Prague
  - PV-Medical s.r.o., Zlín
- Estonia (2):
  - East Tallinn Central Hospital, Tallinn
  - North Estonia Regional Hospital, Tallinn
- India (6):
  - Department of Rheumatology, CARE Hospital, Hyderabad, Andhra Pradesh
  - Nizam's Institute of Medical Sciences, Department of Rheumatology, Hyderabad, Andhra Pradesh
  - St. John's Medical College Hospital, Department of Orthopedics, Bangalore, Karnataka
  - T. N. Medical College and B. Y. L. Nair Ch. HospitalDepartment of Medicine and Rheumatology Clinic, Mumbai, Maharashtra
  - Dayanand Medical College and Hospital, Department of Orthopedics, Ludhiana, Punjab
  - Kovai Medical Center and Hospital,, Coimbatore, Tamil Nadu
- Peru (3):
  - Instituto Peruano del Hueso y la Articulación SAC., Lima
  - Instituto Peruano del Climaterio, Lima
  - Instituto de Ginecologia y Reproduccion, Lima
- Poland (4):
  - SP ZOZ Wojewodzki Szpital Zespolony im. Jedrzeja Sniadeckiego, Bialystok
  - Centrum Osteoporozy i Chorob Kostno-Stawowych, Bialystok
  - Poznanski Osrodek Medyczny, Poznan
  - Centrum Badan Klinicznych, Warsaw
- Russia (5):
  - City Hospital #4, Department of Therapy of Moscow Faculty of Russian State Medical University, Moscow
  - Clinical Hospital #7, Moscow
  - City Hospital # 28 "Maximilianovskaya", Saint Petersburg
  - St. Petersburg Clnical Hospital n.a. Sokolov (MSCh #122), Saint Petersburg
  - Smolensk State Medical Academy, Smolensk
- South Africa (6):
  - Office Of Dr. F. Le Clus, Johannesburg, Gauteng
  - Dr S Sankovic, Parktown, Johannesburg
  - Quinta-Med, Bloemfontein
  - St Augustines Medical Ctr 2, Durban
  - Clinresco Centres (Pty) Ltd, Kempton Park
  - Intercare Medical and Dental Centre, Pretoria
- South Korea (4):
  - Hallym University Sacred Heart Hospital/Rheumatology, Internal Medicine, Anyang
  - Yonsei University College of Medicine, Severance Hospital, Rheumatology, Internal Medicine, Seoul
  - Hanyang University Hospital, Department of Rheumatology, Seoul
  - The Catholic University of Korea, Kangnam St. Mary's Hospital/ Rheumatology, Internal Medicine, Seoul
- Spain (2):
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital Nuestra Señora de Valme, Seville

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6631007&StudyName=An%20Oral%20p38%20Inhibitor%20Investigating%20Safety%2C%20Efficacy%2C%20And%20PK%20In%20Subjects%20With%20Active%20Rheumatoid%20Arthritis

RESULTS

PARTICIPANT FLOW:
Groups:
- PH-797804, 0.5 mg: Participants received PH-797804, 0.5 milligram (mg) capsule, orally, once daily for 12 weeks. Participants were followed up to 28 days after last dose of study drug. Individual participant participated in the study for a duration of up to 16 weeks.
- PH79804, 3 mg: Participants received PH-797804, 3 mg capsule, orally, once daily for 12 weeks. Participants were followed up to 28 days after last dose of study drug. Individual participant participated in the study for a duration of up to 16 weeks.
- PH-797804, 6 mg: Participants received PH-797804, 6 mg capsule, orally, once daily for 12 weeks. Participants were followed up to 28 days after last dose of study drug. Individual participant participated in the study for a duration of up to 16 weeks.
- PH-797804, 10 mg: Participants received PH-797804, 10 mg capsule, orally, once daily for 12 weeks. Participants were followed up to 28 days after last dose of study drug. Individual participant participated in the study for a duration of up to 16 weeks.
- Placebo: Participants received placebo matched to PH-797804, orally, once daily for 12 weeks. Participants were followed up to 28 days after last dose of study drug. Individual participant participated in the study for a duration of up to 16 weeks.
Period: Overall Study
Arm/Group | PH-797804, 0.5 mg | PH79804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Started | 69 | 74 | 44 | 40 | 75
Completed | 52 | 63 | 31 | 28 | 52
Not Completed | 17 | 11 | 13 | 12 | 23
Not completed — Adverse Event | 4 | 7 | 9 | 8 | 8
Not completed — Lack of Efficacy | 9 | 3 | 3 | 2 | 6
Not completed — Other | 3 | 1 | 0 | 2 | 6
Not completed — No longer willing to participate | 1 | 0 | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants randomized to treatment and who had taken at least 1 dose of study medication.
Groups:
- PH-797804, 0.5 mg: Participants received PH-797804, 0.5 mg capsule, orally, once daily for 12 weeks. Participants were followed up to 28 days after last dose of study drug. Individual participant participated in the study for a duration of up to 16 weeks.
- Total: Total of all reporting groups
Arm/Group | PH-797804, 0.5 mg | PH79804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo | Total
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75 | 302
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 59 | 60 | 39 | 36 | 65 | 259
  >=65 years | 10 | 14 | 5 | 4 | 10 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 62 | 38 | 35 | 60 | 256
  Male | 8 | 12 | 6 | 5 | 15 | 46

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20 Percent (%) (ACR 20) Response at Week 12
Description: ACR20 responders: participants with greater than or equal to(>=)20% improvement in tender and swollen 28-joint counts from baseline, >=20% improvement in at least 3 of 5 measures: Patient's global assessment of arthritis(PGA), physician's global assessment of arthritis, participant's assessment of pain on visual analogue scale (Pain-VAS), health assessment questionnaire-disability index (HAQ-DI), C-reactive protein (CRP) in mg/liter (mg/L). PGA:participant assess overall disease activity on VAS, score:0(no arthritis) to 100(extreme arthritis), high score=more arthritis. Physician's global assessment:physician judge participant's overall disease activity on VAS, score:0(no arthritis) to 100millimeter(mm) (extreme arthritis), high score=more arthritis. Pain-VAS:participant assess arthritis pain on 100mm VAS, score:0mm (no pain) to 100mm (extreme pain), high score=more pain. HAQ-DI:functional disability evaluation, score:0 (no difficulty) to 3 (unable to do), high score=more disability.
Time Frame: Week 12
Population: FAS included all participants randomized to treatment and who had taken at least 1 dose of study medication. Here 'overall number of participants analyzed' signifies participants who were evaluable for this outcome measure. Missing values were imputed using last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Groups:
- PH-797804, 3 mg: Participants received PH-797804, 3 mg capsule, orally, once daily for 12 weeks. Participants were followed up to 28 days after last dose of study drug. Individual participant participated in the study for a duration of up to 16 weeks.
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
percentage of participants | 39.13 | 41.89 | 40.91 | 40.00 | 31.08
Statistical Analysis 1: Comparison: PH-797804, 0.5 mg vs Placebo; Test type: Superiority; p = 0.3131, Chi-squared; Difference in percentage = 8.05, 95% CI 2-sided [-7.565 to 23.664], Standard Error of Mean 7.97
Statistical Analysis 2: Comparison: PH-797804, 3 mg vs Placebo; Test type: Superiority; p = 0.1719, Chi-squared; Difference in percentage = 10.81, 95% CI 2-sided [-4.602 to 26.224], Standard Error of Mean 7.86
Statistical Analysis 3: Comparison: PH-797804, 6 mg vs Placebo; Test type: Superiority; p = 0.2783, Chi-squared; Difference in percentage = 9.83, 95% CI 2-sided [-8.123 to 27.799], Standard Error of Mean 9.16
Statistical Analysis 4: Comparison: PH-797804, 10 mg vs Placebo; Test type: Superiority; p = 0.3381, Chi-squared; Difference in percentage = 8.92, 95% CI 2-sided [-9.566 to 27.404], Standard Error of Mean 9.43

2. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20 Percent (%) (ACR 20) Response at Weeks 1, 2, 4, 8 and 16
Description: ACR20 responders: participants with greater than or equal to(>=)20% improvement in tender and swollen 28-joint counts from baseline, >=20% improvement in at least 3 of 5 measures: Patient's global assessment of arthritis(PGA), physician's global assessment of arthritis, participant's assessment of pain on visual analogue scale (Pain-VAS), health assessment questionnaire-disability index (HAQ-DI), C-reactive protein (CRP) in mg/L. PGA:participant assess overall disease activity on VAS, score:0(no arthritis) to 100(extreme arthritis), high score=more arthritis. Physician's global assessment:physician judge participant's overall disease activity on VAS, score:0(no arthritis) to 100millimeter(mm) (extreme arthritis), high score=more arthritis. Pain-VAS:participant assessed arthritis pain on 100mm VAS, score:0mm (no pain) to 100mm (extreme pain), high score=more pain. HAQ-DI:functional disability evaluation, score:0 (no difficulty) to 3 (unable to do), high score=more disability.
Time Frame: Weeks 1, 2, 4, 8, 16
Population: FAS included all participants randomized to treatment and who had taken at least 1 dose of study medication. Here, 'number analyzed' signifies participants evaluable for this outcome measure at specified time points. Missing values were imputed using LOCF except for Week 16.
Measure: Number; unit: percentage of participants
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
percentage of participants
  Week 1: number analyzed (Participants) | 67 | 71 | 43 | 39 | 72
  Week 1 | 14.93 | 21.13 | 27.91 | 15.38 | 13.89
  Week 2: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 2 | 30.43 | 29.73 | 40.91 | 40.00 | 24.32
  Week 4: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 4 | 31.88 | 41.89 | 43.18 | 47.50 | 27.03
  Week 8: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 8 | 28.99 | 45.95 | 40.91 | 47.50 | 31.08
  Week 16: number analyzed (Participants) | 62 | 70 | 38 | 38 | 70
  Week 16 | 38.71 | 42.86 | 44.74 | 28.95 | 41.43
Statistical Analysis 1: Comparison: PH-797804, 0.5 mg vs Placebo; Week 1; Test type: Superiority; p = 0.8619, Chi-squared; Difference in percentage = 1.04, 90% CI 2-sided [-8.733 to 10.845], Standard Error of Mean 5.96
Statistical Analysis 2: Comparison: PH-797804, 3 mg vs Placebo; Week 1; Test type: Superiority; p = 0.2546, Chi-squared; Difference in percentage = 7.24, 90% CI 2-sided [-3.176 to 17.651], Standard Error of Mean 6.33
Statistical Analysis 3: Comparison: PH-797804, 6 mg vs Placebo; Week 1; Test type: Superiority; p = 0.0644, Chi-squared; Difference in percentage = 14.02, 90% CI 2-sided [0.921 to 27.115], Standard Error of Mean 7.96
Statistical Analysis 4: Comparison: PH-797804, 10 mg vs Placebo; Week 1; Test type: Superiority; p = 0.8304, Chi-squared; Difference in percentage = 1.50, 90% CI 2-sided [-10.13 to 13.125], Standard Error of Mean 7.07
Statistical Analysis 5: Comparison: PH-797804, 0.5 mg vs Placebo; Week 2; Test type: Superiority; p = 0.4123, Chi-squared; Difference in percentage = 6.11, 90% CI 2-sided [-6.150 to 18.371], Standard Error of Mean 7.45
Statistical Analysis 6: Comparison: PH-797804, 3 mg vs Placebo; Week 2; Test type: Superiority; p = 0.4591, Chi-squared; Difference in percentage = 5.41, 90% CI 2-sided [-6.581 to 17.392], Standard Error of Mean 7.29
Statistical Analysis 7: Comparison: PH-797804, 6 mg vs Placebo; Week 2; Test type: Superiority; p = 0.0585, Chi-squared; Difference in percentage = 16.58, 90% CI 2-sided [1.890 to 31.280], Standard Error of Mean 8.93
Statistical Analysis 8: Comparison: PH-797804, 10 mg vs Placebo; Week 2; Test type: Superiority; p = 0.0808, Chi-squared; Difference in percentage = 15.68, 90% CI 2-sided [0.522 to 30.829], Standard Error of Mean 9.21
Statistical Analysis 9: Comparison: PH-797804, 0.5 mg vs Placebo; Week 4; Test type: Superiority; p = 0.5240, Chi-squared; Difference in percentage = 4.86, 90% CI 2-sided [-7.684 to 17.398], Standard Error of Mean 7.62
Statistical Analysis 10: Comparison: PH-797804, 3 mg vs Placebo; Week 4; Test type: Superiority; p = 0.0571, Chi-squared; Difference in percentage = 14.86, 90% CI 2-sided [2.172 to 27.588], Standard Error of Mean 7.72
Statistical Analysis 11: Comparison: PH-797804, 6 mg vs Placebo; Week 4; Test type: Superiority; p = 0.0712, Chi-squared; Difference in percentage = 16.15, 90% CI 2-sided [1.222 to 31.087], Standard Error of Mean 9.08
Statistical Analysis 12: Comparison: PH-797804, 10 mg vs Placebo; Week 4; Test type: Superiority; p = 0.0279, Chi-squared; Difference in percentage = 20.47, 90% CI 2-sided [4.956 to 35.990], Standard Error of Mean 9.43
Statistical Analysis 13: Comparison: PH-797804, 0.5 mg vs Placebo; Week 8; Test type: Superiority; p = 0.7848, Chi-squared; Difference in Percentage = -2.10, 90% CI 2-sided [-14.71 to 10.515], Standard Error of Mean 7.67
Statistical Analysis 14: Comparison: PH-797804, 3 mg vs Placebo; Week 8; Test type: Superiority; p = 0.0632, Chi-squared; Difference in percentage = 14.86, 90% CI 2-sided [1.860 to 27.869], Standard Error of Mean 7.91
Statistical Analysis 15: Comparison: PH-797804, 6 mg vs Placebo; Week 8; Test type: Superiority; p = 0.2783, Chi-squared; Difference in percentage = 9.83, 90% CI 2-sided [-5.237 to 24.893], Standard Error of Mean 9.16
Statistical Analysis 16: Comparison: PH-797804, 10 mg vs Placebo; Week 8; Test type: Superiority; p = 0.0828, Chi-squared; Difference in percentage = 16.42, 90% CI 2-sided [0.703 to 32.135], Standard Error of Mean 9.55
Statistical Analysis 17: Comparison: PH-797804, 0.5 mg vs Placebo; Week 16; Test type: Superiority; p = 0.7505, Chi-squared; Difference in percentage = -2.72, 90% CI 2-sided [-16.77 to 11.328], Standard Error of Mean 8.54
Statistical Analysis 18: Comparison: PH-797804, 3 mg vs Placebo; Week 16; Test type: Superiority; p = 0.8641, Chi-squared; Difference in percentage = 1.43, 90% CI 2-sided [-12.30 to 15.156], Standard Error of Mean 8.35
Statistical Analysis 19: Comparison: PH-797804, 6 mg vs Placebo; Week 16; Test type: Superiority; p = 0.7399, Chi-squared; Difference in percentage = 3.31, 90% CI 2-sided [-13.12 to 19.734], Standard Error of Mean 9.99
Statistical Analysis 20: Comparison: PH-797804, 10 mg vs Placebo; Week 16; Test type: Superiority; p = 0.1996, Chi-squared; Difference in percentage = -12.48, 90% CI 2-sided [-27.98 to 3.018], Standard Error of Mean 9.42

3. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50 Percent (%) (ACR 50) Response at Weeks 1, 2, 4, 8, 12 and 16
Description: ACR50 responders: participants with >= 50% improvement in tender and swollen 28-joint counts from baseline and >= 50% improvement in at least 3 of the 5 measures: PGA, physician global assessment, Pain-VAS, HAQ-DI and C-reactive protein (in mg/L). PGA: participant assessed overall disease activity on VAS, score: 0 (no arthritis) to 100 (extreme arthritis), higher score=more arthritis. Physician global assessment: physician judged participant's overall disease activity on VAS, score: 0 (no arthritis) to 100 mm VAS (extreme arthritis), higher score=more arthritis. Pain-VAS: participant assessed arthritis pain by 100 mm VAS, score: 0 mm (no pain) to 100 mm (extreme pain), higher score=more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (unable to do), higher score=more disability.
Time Frame: Weeks 1, 2, 4, 8, 12 and 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
percentage of participants
  Week 1: number analyzed (Participants) | 67 | 71 | 43 | 39 | 72
  Week 1 | 1.49 | 1.41 | 4.65 | 5.13 | 0.00
  Week 2: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 2 | 5.80 | 9.46 | 11.36 | 12.50 | 1.35
  Week 4: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 4 | 2.90 | 13.51 | 18.18 | 17.50 | 5.41
  Week 8: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 8 | 4.35 | 17.57 | 20.45 | 15.00 | 13.51
  Week 12: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 12 | 17.39 | 21.62 | 20.45 | 17.50 | 12.16
  Week 16: number analyzed (Participants) | 62 | 70 | 38 | 38 | 70
  Week 16 | 19.35 | 18.57 | 15.79 | 5.26 | 21.43
Statistical Analysis 1: Comparison: PH-797804, 0.5 mg vs Placebo; Week 1; Test type: Superiority; p = 0.2982, Chi-squared; Difference in percentage = 1.49, 90% CI 2-sided [-0.944 to 3.929], Standard Error of Mean 1.48
Statistical Analysis 2: Comparison: PH-797804, 3 mg vs Placebo; Week 1; Test type: Superiority; p = 0.3122, Chi-squared; Difference in percentage = 1.41, 90% CI 2-sided [-0.892 to 3.709], Standard Error of Mean 1.40
Statistical Analysis 3: Comparison: PH-797804, 6 mg vs Placebo; Week 1; Test type: Superiority; p = 0.0649, Chi-squared; Difference in percentage = 4.65, 90% CI 2-sided [-0.631 to 9.934], Standard Error of Mean 3.21
Statistical Analysis 4: Comparison: PH-797804, 10 mg vs Placebo; Week 1; Test type: Superiority; p = 0.0525, Chi-squared; Difference in percentage = 5.13, 90% CI 2-sided [-0.681 to 10.938], Standard Error of Mean 3.53
Statistical Analysis 5: Comparison: PH-797804, 0.5 mg vs Placebo; Week 2; Test type: Superiority; p = 0.1481, Chi-squared; Difference in percentage = 4.45, 90% CI 2-sided [-0.681 to 9.573], Standard Error of Mean 3.12
Statistical Analysis 6: Comparison: PH-797804, 3 mg vs Placebo; Week 2; Test type: Superiority; p = 0.0292, Chi-squared; Difference in percentage = 8.11, 90% CI 2-sided [2.093 to 14.124], Standard Error of Mean 3.66
Statistical Analysis 7: Comparison: PH-797804, 6 mg vs Placebo; Week 2; Test type: Superiority; p = 0.0167, Chi-squared; Difference in percentage = 10.01, 90% CI 2-sided [1.839 to 18.186], Standard Error of Mean 4.97
Statistical Analysis 8: Comparison: PH-797804, 10 mg vs Placebo; Week 2; Test type: Superiority; p = 0.0110, Chi-squared; Difference in percentage = 11.15, 90% CI 2-sided [2.269 to 20.029], Standard Error of Mean 5.40
Statistical Analysis 9: Comparison: PH-797804, 0.5 mg vs Placebo; Week 4; Test type: Superiority; p = 0.4550, Chi-squared; Difference in percentage = -2.51, 90% CI 2-sided [-7.959 to 2.946], Standard Error of Mean 3.31
Statistical Analysis 10: Comparison: PH-797804, 3 mg vs Placebo; Week 4; Test type: Superiority; p = 0.0919, Chi-squared; Difference in percentage = 8.11, 90% CI 2-sided [0.271 to 15.946], Standard Error of Mean 4.76
Statistical Analysis 11: Comparison: PH-797804, 6 mg vs Placebo; Week 4; Test type: Superiority; p = 0.0264, Chi-squared; Difference in percentage = 12.78, 90% CI 2-sided [2.280 to 23.272], Standard Error of Mean 6.38
Statistical Analysis 12: Comparison: PH-797804, 10 mg vs Placebo; Week 4; Test type: Superiority; p = 0.0369, Chi-squared; Difference in percentage = 12.09, 90% CI 2-sided [1.308 to 22.881], Standard Error of Mean 6.56
Statistical Analysis 13: Comparison: PH-797804, 0.5 mg vs Placebo; Week 8; Test type: Superiority; p = 0.0568, Chi-squared; Difference in percentage = -9.17, 90% CI 2-sided [-16.85 to -1.482], Standard Error of Mean 4.67
Statistical Analysis 14: Comparison: PH-797804, 3 mg vs Placebo; Week 8; Test type: Superiority; p = 0.4961, Chi-squared; Difference in percentage = 4.05, 90% CI 2-sided [-5.727 to 13.835], Standard Error of Mean 5.95
Statistical Analysis 15: Comparison: PH-797804, 6 mg vs Placebo; Week 8; Test type: Superiority; p = 0.3212, Chi-squared; Difference in percentage = 6.94, 90% CI 2-sided [-5.008 to 18.890], Standard Error of Mean 7.26
Statistical Analysis 16: Comparison: PH-797804, 10 mg vs Placebo; Week 8; Test type: Superiority; p = 0.8274, Chi-squared; Difference in percentage = 1.49, 90% CI 2-sided [-9.870 to 12.843], Standard Error of Mean 6.90
Statistical Analysis 17: Comparison: PH-797804, 0.5 mg vs Placebo; Week 12; Test type: Superiority; p = 0.3774, Chi-squared; Difference in percentage = 5.23, 90% CI 2-sided [-4.538 to 14.996], Standard Error of Mean 5.94
Statistical Analysis 18: Comparison: PH-797804, 3 mg vs Placebo; Week 12; Test type: Superiority; p = 0.1246, Chi-squared; Difference in percentage = 9.46, 90% CI 2-sided [-0.591 to 19.510], Standard Error of Mean 6.11
Statistical Analysis 19: Comparison: PH-797804, 6 mg vs Placebo; Week 12; Test type: Superiority; p = 0.2257, Chi-squared; Difference in percentage = 8.29, 90% CI 2-sided [-3.502 to 20.087], Standard Error of Mean 7.17
Statistical Analysis 20: Comparison: PH-797804, 10 mg vs Placebo; Week 12; Test type: Superiority; p = 0.4336, Chi-squared; Difference in percentage = 5.34, 90% CI 2-sided [-6.355 to 17.030], Standard Error of Mean 7.11
Statistical Analysis 21: Comparison: PH-797804, 0.5 mg vs Placebo; Week 16; Test type: Superiority; p = 0.7682, Chi-squared; Difference in percentage = -2.07, 90% CI 2-sided [-13.61 to 9.467], Standard Error of Mean 7.02
Statistical Analysis 22: Comparison: PH-797804, 3 mg vs Placebo; Week 16; Test type: Superiority; p = 0.6726, Chi-squared; Difference in percentage = -2.86, 90% CI 2-sided [-13.97 to 8.257], Standard Error of Mean 6.76
Statistical Analysis 23: Comparison: PH-797804, 6 mg vs Placebo; Week 16; Test type: Superiority; p = 0.4795, Chi-squared; Difference in percentage = -5.64, 90% CI 2-sided [-18.28 to 7.000], Standard Error of Mean 7.68
Statistical Analysis 24: Comparison: PH-797804, 10 mg vs Placebo; Week 16; Test type: Superiority; p = 0.0276, Chi-squared; Difference in percentage = -16.17, 90% CI 2-sided [-26.19 to -6.137], Standard Error of Mean 6.10

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70 Percent (%) (ACR 70) Response at Weeks 1, 2, 4, 8, 12 and 16
Description: ACR70 responders: participants with >=70% improvement in tender and swollen 28-joint counts from baseline and >= 70% improvement in at least 3 of the 5 measures: PGA, physician global assessment, Pain-VAS, HAQ-DI and CRP (in mg/L). PGA: participant assessed overall disease activity on VAS, score: 0 (no arthritis) to 100 (extreme arthritis), higher score=more arthritis. Physician global assessment: physician judged participant's overall disease activity on VAS, score: 0 (no arthritis) to 100 mm VAS (extreme arthritis), higher score=more arthritis. Pain-VAS: participant assessed arthritis pain by 100 mm VAS, score: 0 mm (no pain) to 100 mm (extreme pain), higher score=more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (unable to do), higher score=more disability.
Time Frame: Weeks 1, 2, 4, 8, 12 and 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
percentage of participants
  Week 1: number analyzed (Participants) | 67 | 71 | 43 | 39 | 72
  Week 1 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Week 2: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 2 | 0.00 | 0.00 | 2.27 | 2.50 | 0.00
  Week 4: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 4 | 1.45 | 0.00 | 6.82 | 5.00 | 1.35
  Week 8: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 8 | 1.45 | 4.05 | 11.36 | 10.00 | 4.05
  Week 12: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 12 | 7.25 | 8.11 | 9.09 | 7.50 | 5.41
  Week 16: number analyzed (Participants) | 62 | 70 | 38 | 38 | 70
  Week 16 | 4.84 | 7.14 | 2.63 | 2.63 | 10.00
Statistical Analysis 1: Comparison: PH-797804, 0.5 mg vs Placebo; Week 1; Test type: Superiority; p = 0.000, Chi-squared; Difference in percentage = 0.00, 90% CI 2-sided [0.00 to 0.00], Standard Error of Mean 0.00
Statistical Analysis 2: Comparison: PH-797804, 3 mg vs Placebo; Week 1; Test type: Superiority; p = 0.000, Chi-squared; Difference in percentage = 0.00, 90% CI 2-sided [0.00 to 0.00], Standard Error of Mean 0.00
Statistical Analysis 3: Comparison: PH-797804, 6 mg vs Placebo; Week 1; Test type: Superiority; p = 0.000, Chi-squared; Difference in percentage = 0.00, 90% CI 2-sided [0.00 to 0.00], Standard Error of Mean 0.00
Statistical Analysis 4: Comparison: PH-797804, 10 mg vs Placebo; Week 1; Test type: Superiority; p = 0.000, Chi-squared; Difference in percentage = 0.00, 90% CI 2-sided [0.00 to 0.00], Standard Error of Mean 0.00
Statistical Analysis 5: Comparison: PH-797804, 0.5 mg vs Placebo; Week 2; Test type: Superiority; p = 0.000, Chi-squared; Difference in percentage = 0.00, 90% CI 2-sided [0.00 to 0.00], Standard Error of Mean 0.00
Statistical Analysis 6: Comparison: PH-797804, 3 mg vs Placebo; Week 2; Test type: Superiority; p = 0.000, Chi-squared; Difference in percentage = 0.00, 90% CI 2-sided [0.00 to 0.00], Standard Error of Mean 0.00
Statistical Analysis 7: Comparison: PH-797804, 6 mg vs Placebo; Week 2; Test type: Superiority; p = 0.1928, Chi-squared; Difference in percentage = 2.27, 90% CI 2-sided [-1.423 to 5.968], Standard Error of Mean 2.25
Statistical Analysis 8: Comparison: PH-797804, 10 mg vs Placebo; Week 2; Test type: Superiority; p = 0.1719, Chi-squared; Difference in percentage = 2.50, 90% CI 2-sided [-1.560 to 6.560], Standard Error of Mean 2.47
Statistical Analysis 9: Comparison: PH-797804, 0.5 mg vs Placebo; Week 4; Test type: Superiority; p = 0.9603, Chi-squared; Difference in percentage = 0.10, 90% CI 2-sided [-3.138 to 3.334], Standard Error of Mean 1.97
Statistical Analysis 10: Comparison: PH-797804, 3 mg vs Placebo; Week 4; Test type: Superiority; p = 0.3157, Chi-squared; Difference in percentage = -1.35, 90% CI 2-sided [-3.559 to 0.856], Standard Error of Mean 1.34
Statistical Analysis 11: Comparison: PH-797804, 6 mg vs Placebo; Week 4; Test type: Superiority; p = 0.1125, Chi-squared; Difference in percentage = 5.47, 90% CI 2-sided [-1.162 to 12.096], Standard Error of Mean 4.03
Statistical Analysis 12: Comparison: PH-797804, 10 mg vs Placebo; Week 4; Test type: Superiority; p = 0.2455, Chi-squared; Difference in percentage = 3.65, 90% CI 2-sided [-2.434 to 9.732], Standard Error of Mean 3.70
Statistical Analysis 13: Comparison: PH-797804, 0.5 mg vs Placebo; Week 8; Test type: Superiority; p = 0.3452, Chi-squared; Difference in percentage = -2.60, 90% CI 2-sided [-7.057 to 1.847], Standard Error of Mean 2.71
Statistical Analysis 14: Comparison: PH-797804, 3 mg vs Placebo; Week 8; Test type: Superiority; p = 1.0000, Chi-squared; Difference in percentage = 0.00, 90% CI 2-sided [-5.333 to 5.333], Standard Error of Mean 3.24
Statistical Analysis 15: Comparison: PH-797804, 6 mg vs Placebo; Week 8; Test type: Superiority; p = 0.1267, Chi-squared; Difference in percentage = 7.31, 90% CI 2-sided [-1.417 to 16.036], Standard Error of Mean 5.31
Statistical Analysis 16: Comparison: PH-797804, 10 mg vs Placebo; Week 8; Test type: Superiority; p = 0.2069, Chi-squared; Difference in percentage = 5.95, 90% CI 2-sided [-2.720 to 14.612], Standard Error of Mean 5.27
Statistical Analysis 17: Comparison: PH-797804, 0.5 mg vs Placebo; Week 12; Test type: Superiority; p = 0.6506, Chi-squared; Difference in percentage = 1.84, 90% CI 2-sided [-4.871 to 8.553], Standard Error of Mean 4.08
Statistical Analysis 18: Comparison: PH-797804, 3 mg vs Placebo; Week 12; Test type: Superiority; p = 0.5125, Chi-squared; Difference in percentage = 2.70, 90% CI 2-sided [-4.075 to 9.480], Standard Error of Mean 4.12
Statistical Analysis 19: Comparison: PH-797804, 6 mg vs Placebo; Week 12; Test type: Superiority; p = 0.4412, Chi-squared; Difference in percentage = 3.69, 90% CI 2-sided [-4.652 to 12.023], Standard Error of Mean 5.07
Statistical Analysis 20: Comparison: PH-797804, 10 mg vs Placebo; Week 12; Test type: Superiority; p = 0.6566, Chi-squared; Difference in percentage = 2.09, 90% CI 2-sided [-6.006 to 10.195], Standard Error of Mean 4.92
Statistical Analysis 21: Comparison: PH-797804, 0.5 mg vs Placebo; Week 16; Test type: Superiority; p = 0.2634, Chi-squared; Difference in percentage = -5.16, 90% CI 2-sided [-12.57 to 2.247], Standard Error of Mean 4.50
Statistical Analysis 22: Comparison: PH-797804, 3 mg vs Placebo; Week 16; Test type: Superiority; p = 0.5460, Chi-squared; Difference in percentage = -2.86, 90% CI 2-sided [-10.63 to 4.916], Standard Error of Mean 4.73
Statistical Analysis 23: Comparison: PH-797804, 6 mg vs Placebo; Week 16; Test type: Superiority; p = 0.1626, Chi-squared; Difference in percentage = -7.37, 90% CI 2-sided [-14.65 to -0.086], Standard Error of Mean 4.43
Statistical Analysis 24: Comparison: PH-797804, 10 mg vs Placebo; Week 16; Test type: Superiority; p = 0.1626, Chi-squared; Difference in percentage = -7.37, 90% CI 2-sided [-14.65 to -0.086], Standard Error of Mean 4.43

5. Secondary Outcome: Change From Baseline in Tender/Painful Joint Count at Weeks 1, 2, 4, 8, 12 and 16
Description: A total of 28 tender/painful joints were assessed for tenderness or pain. The 28 joints included: shoulders, elbows, wrists, metacarpophalangeal (MCP) joints, proximal interphalangeal (PIP) joints, and knees. Artificial joints were not assessed.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12 and 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Joint count
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
Joint count
  Week 1: number analyzed (Participants) | 67 | 71 | 43 | 39 | 72
  Week 1 | -2.486 (0.751) | -3.409 (0.722) | -4.285 (0.944) | -2.948 (0.981) | -2.098 (0.730)
  Week 2: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 2 | -4.291 (0.746) | -4.334 (0.714) | -5.751 (0.938) | -4.348 (0.975) | -3.003 (0.724)
  Week 4: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 4 | -5.132 (0.746) | -4.982 (0.714) | -5.774 (0.938) | -4.723 (0.975) | -3.368 (0.724)
  Week 8: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 8 | -4.827 (0.746) | -6.090 (0.714) | -5.797 (0.938) | -5.223 (0.975) | -4.069 (0.723)
  Week 12: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 12 | -5.842 (0.746) | -5.996 (0.714) | -6.146 (0.938) | -5.673 (0.975) | -3.762 (0.722)
  Week 16: number analyzed (Participants) | 60 | 70 | 38 | 35 | 68
  Week 16 | -5.505 (0.776) | -4.982 (0.725) | -5.560 (0.977) | -5.069 (1.011) | -5.254 (0.738)
Statistical Analysis 1: Comparison: PH-797804, 0.5 mg vs Placebo; Week 1: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 1 as an interaction term, baseline tender/ joint count as the covariate and participant as a random effect; Test type: Superiority; p = 0.7053, ANCOVA; Least Square Mean (LSM) Difference = -0.388, 95% CI 2-sided [-2.400 to 1.624], Standard Error of Mean 1.025
Statistical Analysis 2: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.1938, ANCOVA; LSM Difference = -1.312, 95% CI 2-sided [-3.291 to 0.668], Standard Error of Mean 1.009
Statistical Analysis 3: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0627, ANCOVA; LSM Difference = -2.187, 95% CI 2-sided [-4.491 to 0.116], Standard Error of Mean 1.174
Statistical Analysis 4: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.4809, ANCOVA; LSM Difference = -0.851, 95% CI 2-sided [-3.218 to 1.517], Standard Error of Mean 1.206
Statistical Analysis 5: Comparison: PH-797804, 0.5 mg vs Placebo; Week 2: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 2 as an interaction term, baseline tender/ joint count as the covariate and participant as a random effect; Test type: Superiority; p = 0.2057, ANCOVA; LSM Difference = -1.289, 95% CI 2-sided [-3.286 to 0.709], Standard Error of Mean 1.017
Statistical Analysis 6: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.1833, ANCOVA; LSM Difference = -1.331, 95% CI 2-sided [-3.293 to 0.631], Standard Error of Mean 0.999
Statistical Analysis 7: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.0187, ANCOVA; LSM Difference = -2.748, 95% CI 2-sided [-5.037 to -0.459], Standard Error of Mean 1.166
Statistical Analysis 8: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.2615, ANCOVA; LSM Difference = -1.345, 95% CI 2-sided [-3.695 to 1.005], Standard Error of Mean 1.197
Statistical Analysis 9: Comparison: PH-797804, 0.5 mg vs Placebo; Week 4: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 4 as an interaction term, baseline tender/ joint count as the covariate and participant as a random effect; Test type: Superiority; p = 0.0832, ANCOVA; LSM Difference = -1.764, 95% CI 2-sided [-3.761 to 0.233], Standard Error of Mean 1.017
Statistical Analysis 10: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 5, analysis 9]; Test type: Superiority; p = 0.1066, ANCOVA; LSM Difference = -1.615, 95% CI 2-sided [-3.576 to 0.347], Standard Error of Mean 0.999
Statistical Analysis 11: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 5, analysis 9]; Test type: Superiority; p = 0.0394, ANCOVA; LSM Difference = -2.406, 95% CI 2-sided [-4.695 to -0.118], Standard Error of Mean 1.166
Statistical Analysis 12: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 5, analysis 9]; Test type: Superiority; p = 0.2580, ANCOVA; LSM Difference = -1.355, 95% CI 2-sided [-3.705 to 0.995], Standard Error of Mean 1.197
Statistical Analysis 13: Comparison: PH-797804, 0.5 mg vs Placebo; Week 8: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 8 as an interaction term, baseline tender/ joint count as the covariate and participant as a random effect; Test type: Superiority; p = 0.4560, ANCOVA; LSM Difference = -0.758, 95% CI 2-sided [-2.754 to 1.238], Standard Error of Mean 1.017
Statistical Analysis 14: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 5, analysis 13]; Test type: Superiority; p = 0.0434, ANCOVA; LSM Difference = -2.021, 95% CI 2-sided [-3.982 to -0.060], Standard Error of Mean 0.999
Statistical Analysis 15: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 5, analysis 13]; Test type: Superiority; p = 0.1386, ANCOVA; LSM Difference = -1.728, 95% CI 2-sided [-4.016 to 0.560], Standard Error of Mean 1.165
Statistical Analysis 16: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 5, analysis 13]; Test type: Superiority; p = 0.3353, ANCOVA; LSM Difference = -1.154, 95% CI 2-sided [-3.503 to 1.196], Standard Error of Mean 1.197
Statistical Analysis 17: Comparison: PH-797804, 0.5 mg vs Placebo; Week 12: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 12 as an interaction term, baseline tender/ joint count as the covariate and participant as a random effect; Test type: Superiority; p = 0.0410, ANCOVA; LSM Difference = -2.080, 95% CI 2-sided [-4.075 to -0.085], Standard Error of Mean 1.016
Statistical Analysis 18: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 5, analysis 17]; Test type: Superiority; p = 0.0255, ANCOVA; LSM Difference = -2.234, 95% CI 2-sided [-4.194 to -0.274], Standard Error of Mean 0.998
Statistical Analysis 19: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 5, analysis 17]; Test type: Superiority; p = 0.0410, ANCOVA; LSM Difference = -2.384, 95% CI 2-sided [-4.671 to -0.097], Standard Error of Mean 1.165
Statistical Analysis 20: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 5, analysis 17]; Test type: Superiority; p = 0.1106, ANCOVA; LSM Difference = -1.911, 95% CI 2-sided [-4.259 to 0.438], Standard Error of Mean 1.196
Statistical Analysis 21: Comparison: PH-797804, 0.5 mg vs Placebo; Week 16: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 16 as an interaction term, baseline tender/ joint count as the covariate and participant as a random effect; Test type: Superiority; p = 0.8107, ANCOVA; LSM Difference = -0.251, 95% CI 2-sided [-2.307 to 1.805], Standard Error of Mean 1.048
Statistical Analysis 22: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 5, analysis 21]; Test type: Superiority; p = 0.7895, ANCOVA; LSM Difference = 0.272, 95% CI 2-sided [-1.726 to 2.269], Standard Error of Mean 1.017
Statistical Analysis 23: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 5, analysis 21]; Test type: Superiority; p = 0.7996, ANCOVA; LSM Difference = -0.306, 95% CI 2-sided [-2.673 to 2.060], Standard Error of Mean 1.206
Statistical Analysis 24: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 5, analysis 21]; Test type: Superiority; p = 0.8811, ANCOVA; LSM Difference = 0.185, 95% CI 2-sided [-2.240 to 2.610], Standard Error of Mean 1.235

6. Secondary Outcome: Change From Baseline in Swollen Joint Count at Weeks 1, 2, 4, 8, 12 and 16
Description: A total of 28 swollen joints were assessed. The 28 joints included: shoulders, elbows, wrists, MCP joints, PIP joints, and knees. Artificial joints were not assessed.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12 and 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Joint count
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
Joint count
  Week 1: number analyzed (Participants) | 67 | 71 | 43 | 39 | 72
  Week 1 | -2.341 (0.650) | -2.738 (0.625) | -3.224 (0.816) | -2.328 (0.849) | -1.654 (0.633)
  Week 2: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 2 | -3.847 (0.645) | -3.409 (0.618) | -4.041 (0.811) | -3.187 (0.843) | -2.382 (0.629)
  Week 4: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 4 | -4.368 (0.645) | -4.369 (0.618) | -4.599 (0.811) | -3.262 (0.843) | -2.769 (0.628)
  Week 8: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 8 | -4.412 (0.645) | -4.504 (0.618) | -4.134 (0.811) | -3.937 (0.843) | -3.236 (0.628)
  Week 12: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 12 | -4.992 (0.645) | -4.477 (0.618) | -4.227 (0.811) | -3.587 (0.843) | -3.391 (0.627)
  Week 16: number analyzed (Participants) | 60 | 70 | 38 | 35 | 68
  Week 16 | -4.300 (0.669) | -4.168 (0.626) | -4.138 (0.842) | -4.166 (0.872) | -4.676 (0.640)
Statistical Analysis 1: Comparison: PH-797804, 0.5 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.4385, ANCOVA; LSM Difference = -0.687, 95% CI 2-sided [-2.427 to 1.053], Standard Error of Mean 0.886
Statistical Analysis 2: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.2131, ANCOVA; LSM Difference = -1.085, 95% CI 2-sided [-2.794 to 0.624], Standard Error of Mean 0.870
Statistical Analysis 3: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.1216, ANCOVA; LSM Difference = -1.570, 95% CI 2-sided [-3.559 to 0.419], Standard Error of Mean 1.013
Statistical Analysis 4: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.5190, ANCOVA; LSM Difference = -0.675, 95% CI 2-sided [-2.728 to 1.378], Standard Error of Mean 1.046
Statistical Analysis 5: Comparison: PH-797804, 0.5 mg vs Placebo; Week 2: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 2 as an interaction term, baseline swollen joint count as the covariate and participant as a random effect; Test type: Superiority; p = 0.0967, ANCOVA; LSM Difference = -1.464, 95% CI 2-sided [-3.193 to 0.264], Standard Error of Mean 0.880
Statistical Analysis 6: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 6, analysis 5]; Test type: Superiority; p = 0.2346, ANCOVA; LSM Difference = -1.027, 95% CI 2-sided [-2.721 to 0.668], Standard Error of Mean 0.863
Statistical Analysis 7: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 6, analysis 5]; Test type: Superiority; p = 0.1000, ANCOVA; LSM Difference = -1.658, 95% CI 2-sided [-3.635 to 0.318], Standard Error of Mean 1.007
Statistical Analysis 8: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 6, analysis 5]; Test type: Superiority; p = 0.4385, ANCOVA; LSM Difference = -0.805, 95% CI 2-sided [-2.844 to 1.234], Standard Error of Mean 1.038
Statistical Analysis 9: Comparison: PH-797804, 0.5 mg vs Placebo; Week 4: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 4 as an interaction term, baseline swollen joint count as the covariate and participant as a random effect; Test type: Superiority; p = 0.0696, ANCOVA; LSM Difference = -1.599, 95% CI 2-sided [-3.327 to 0.128], Standard Error of Mean 0.880
Statistical Analysis 10: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 6, analysis 9]; Test type: Superiority; p = 0.0642, ANCOVA; LSM Difference = -1.600, 95% CI 2-sided [-3.294 to 0.094], Standard Error of Mean 0.863
Statistical Analysis 11: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 6, analysis 9]; Test type: Superiority; p = 0.0695, ANCOVA; LSM Difference = -1.830, 95% CI 2-sided [-3.807 to 0.146], Standard Error of Mean 1.007
Statistical Analysis 12: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 6, analysis 9]; Test type: Superiority; p = 0.6349, ANCOVA; LSM Difference = -0.493, 95% CI 2-sided [-2.532 to 1.545], Standard Error of Mean 1.038
Statistical Analysis 13: Comparison: PH-797804, 0.5 mg vs Placebo; Week 8: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 8 as an interaction term, baseline swollen joint count as the covariate and participant as a random effect; Test type: Superiority; p = 0.1818, ANCOVA; LSM Difference = -1.176, 95% CI 2-sided [-2.903 to 0.551], Standard Error of Mean 0.880
Statistical Analysis 14: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority; p = 0.1421, ANCOVA; LSM Difference = -1.268, 95% CI 2-sided [-2.961 to 0.426], Standard Error of Mean 0.862
Statistical Analysis 15: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority; p = 0.3726, ANCOVA; LSM Difference = -0.898, 95% CI 2-sided [-2.874 to 1.078], Standard Error of Mean 1.006
Statistical Analysis 16: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority; p = 0.4995, ANCOVA; LSM Difference = -0.701, 95% CI 2-sided [-2.739 to 1.337], Standard Error of Mean 1.038
Statistical Analysis 17: Comparison: PH-797804, 0.5 mg vs Placebo; Week 12: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 12 as an interaction term, baseline swollen joint count as the covariate and participant as a random effect; Test type: Superiority; p = 0.0691, ANCOVA; LSM Difference = -1.601, 95% CI 2-sided [-3.327 to 0.126], Standard Error of Mean 0.879
Statistical Analysis 18: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 6, analysis 17]; Test type: Superiority; p = 0.2083, ANCOVA; LSM Difference = -1.086, 95% CI 2-sided [-2.778 to 0.607], Standard Error of Mean 0.862
Statistical Analysis 19: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 6, analysis 17]; Test type: Superiority; p = 0.4063, ANCOVA; LSM Difference = -0.836, 95% CI 2-sided [-2.811 to 1.139], Standard Error of Mean 1.006
Statistical Analysis 20: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 6, analysis 17]; Test type: Superiority; p = 0.8501, ANCOVA; LSM Difference = -0.196, 95% CI 2-sided [-2.234 to 1.841], Standard Error of Mean 1.038
Statistical Analysis 21: Comparison: PH-797804, 0.5 mg vs Placebo; Week 16: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 16 as an interaction term, baseline swollen joint count as the covariate and participant as a random effect; Test type: Superiority; p = 0.6778, ANCOVA; LSM Difference = 0.376, 95% CI 2-sided [-1.399 to 2.150], Standard Error of Mean 0.904
Statistical Analysis 22: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 6, analysis 21]; Test type: Superiority; p = 0.5627, ANCOVA; LSM Difference = 0.508, 95% CI 2-sided [-1.214 to 2.230], Standard Error of Mean 0.877
Statistical Analysis 23: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 6, analysis 21]; Test type: Superiority; p = 0.6049, ANCOVA; LSM Difference = 0.537, 95% CI 2-sided [-1.501 to 2.576], Standard Error of Mean 1.038
Statistical Analysis 24: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 6, analysis 21]; Test type: Superiority; p = 0.6332, ANCOVA; LSM Difference = 0.510, 95% CI 2-sided [-1.587 to 2.608], Standard Error of Mean 1.068

7. Secondary Outcome: Change From Baseline in Participant Assessment of Arthritis Pain at Weeks 1, 2, 4, 8, 12 and 16
Description: Participants self-assessed the severity of arthritis pain using a 100 mm VAS between 0 mm (no pain) and 100 mm (most severe pain), where higher scores indicate higher degree of pain intensity.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12 and 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Millimeter (mm)
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
Millimeter (mm)
  Week 1: number analyzed (Participants) | 66 | 71 | 42 | 39 | 72
  Week 1 | -9.289 (3.012) | -16.67 (2.876) | -19.22 (3.796) | -17.62 (3.919) | -6.486 (2.907)
  Week 2: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 2 | -16.50 (2.977) | -19.52 (2.842) | -23.16 (3.746) | -16.93 (3.889) | -9.058 (2.884)
  Week 4: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 4 | -13.82 (2.977) | -21.79 (2.842) | -19.95 (3.746) | -13.76 (3.889) | -11.85 (2.884)
  Week 8: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 8 | -10.86 (2.977) | -23.37 (2.842) | -20.65 (3.746) | -18.68 (3.889) | -12.72 (2.883)
  Week 12: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 12 | -15.06 (2.977) | -21.37 (2.842) | -19.18 (3.746) | -20.38 (3.889) | -10.30 (2.880)
  Week 16: number analyzed (Participants) | 60 | 70 | 38 | 35 | 68
  Week 16 | -14.20 (3.104) | -20.88 (2.888) | -15.19 (3.913) | -14.70 (4.047) | -19.09 (2.949)
Statistical Analysis 1: Comparison: PH-797804, 0.5 mg vs Placebo; Week 1: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 1 as an interaction term, baseline Patient's Assessment of Arthritis Pain (VAS) count as the covariate and participant as a random effect; Test type: Superiority; p = 0.4943, ANCOVA; LSM Difference = -2.802, 95% CI 2-sided [-10.85 to 5.243], Standard Error of Mean 4.098
Statistical Analysis 2: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0116, ANCOVA; LSM Difference = -10.19, 95% CI 2-sided [-18.09 to -2.283], Standard Error of Mean 4.026
Statistical Analysis 3: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0070, ANCOVA; LSM Difference = -12.73, 95% CI 2-sided [-21.98 to -3.485], Standard Error of Mean 4.710
Statistical Analysis 4: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0209, ANCOVA; LSM Difference = -11.14, 95% CI 2-sided [-20.58 to -1.688], Standard Error of Mean 4.812
Statistical Analysis 5: Comparison: PH-797804, 0.5 mg vs Placebo; Week 2:Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 2 as an interaction term, baseline Patient's Assessment of Arthritis Pain (VAS) count as the covariate and participant as a random effect; Test type: Superiority; p = 0.0671, ANCOVA; LSM Difference = -7.439, 95% CI 2-sided [-15.40 to 0.524], Standard Error of Mean 4.056
Statistical Analysis 6: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 7, analysis 5]; Test type: Superiority; p = 0.0089, ANCOVA; LSM Difference = -10.46, 95% CI 2-sided [-18.28 to -2.632], Standard Error of Mean 3.986
Statistical Analysis 7: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 7, analysis 5]; Test type: Superiority; p = 0.0025, ANCOVA; LSM Difference = -14.10, 95% CI 2-sided [-23.24 to -4.959], Standard Error of Mean 4.657
Statistical Analysis 8: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 7, analysis 5]; Test type: Superiority; p = 0.0994, ANCOVA; LSM Difference = -7.876, 95% CI 2-sided [-17.25 to 1.496], Standard Error of Mean 4.774
Statistical Analysis 9: Comparison: PH-797804, 0.5 mg vs Placebo; Week 4: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 4 as an interaction term, baseline Patient's Assessment of Arthritis Pain (VAS) count as the covariate and participant as a random effect; Test type: Superiority; p = 0.6284, ANCOVA; LSM Difference = -1.964, 95% CI 2-sided [-9.926 to 5.999], Standard Error of Mean 4.056
Statistical Analysis 10: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 7, analysis 9]; Test type: Superiority; p = 0.0129, ANCOVA; LSM Difference = -9.934, 95% CI 2-sided [-17.76 to -2.109], Standard Error of Mean 3.986
Statistical Analysis 11: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 7, analysis 9]; Test type: Superiority; p = 0.0825, ANCOVA; LSM Difference = -8.097, 95% CI 2-sided [-17.24 to 1.044], Standard Error of Mean 4.656
Statistical Analysis 12: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 7, analysis 9]; Test type: Superiority; p = 0.6897, ANCOVA; LSM Difference = -1.907, 95% CI 2-sided [-11.28 to 7.465], Standard Error of Mean 4.774
Statistical Analysis 13: Comparison: PH-797804, 0.5 mg vs Placebo; Week 8: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 8 as an interaction term, baseline Patient's Assessment of Arthritis Pain (VAS) count as the covariate and participant as a random effect; Test type: Superiority; p = 0.6465, ANCOVA; LSM Difference = 1.861, 95% CI 2-sided [-6.100 to 9.821], Standard Error of Mean 4.055
Statistical Analysis 14: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority; p = 0.0077, ANCOVA; LSM Difference = -10.65, 95% CI 2-sided [-18.47 to -2.824], Standard Error of Mean 3.985
Statistical Analysis 15: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority; p = 0.0890, ANCOVA; LSM Difference = -7.927, 95% CI 2-sided [-17.07 to 1.213], Standard Error of Mean 4.655
Statistical Analysis 16: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority; p = 0.2119, ANCOVA; LSM Difference = -5.964, 95% CI 2-sided [-15.33 to 3.406], Standard Error of Mean 4.773
Statistical Analysis 17: Comparison: PH-797804, 0.5 mg vs Placebo; Week 12: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 12 as an interaction term, baseline Patient's Assessment of Arthritis Pain (VAS) count as the covariate and participant as a random effect; Test type: Superiority; p = 0.2401, ANCOVA; LSM Difference = -4.766, 95% CI 2-sided [-12.72 to 3.191], Standard Error of Mean 4.053
Statistical Analysis 18: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 7, analysis 17]; Test type: Superiority; p = 0.0056, ANCOVA; LSM Difference = -11.07, 95% CI 2-sided [-18.89 to -3.251], Standard Error of Mean 3.983
Statistical Analysis 19: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 7, analysis 17]; Test type: Superiority; p = 0.0566, ANCOVA; LSM Difference = -8.885, 95% CI 2-sided [-18.02 to 0.251], Standard Error of Mean 4.654
Statistical Analysis 20: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 7, analysis 17]; Test type: Superiority; p = 0.0348, ANCOVA; LSM Difference = -10.09, 95% CI 2-sided [-19.45 to -0.720], Standard Error of Mean 4.772
Statistical Analysis 21: Comparison: PH-797804, 0.5 mg vs Placebo; Week 16: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 16 as an interaction term, baseline Patient's Assessment of Arthritis Pain (VAS) count as the covariate and participant as a random effect; Test type: Superiority; p = 0.2436, ANCOVA; LSM Difference = 4.890, 95% CI 2-sided [-3.336 to 13.116], Standard Error of Mean 4.191
Statistical Analysis 22: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 7, analysis 21]; Test type: Superiority; p = 0.6616, ANCOVA; LSM Difference = -1.781, 95% CI 2-sided [-9.762 to 6.201], Standard Error of Mean 4.066
Statistical Analysis 23: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 7, analysis 21]; Test type: Superiority; p = 0.4189, ANCOVA; LSM Difference = 3.907, 95% CI 2-sided [-5.574 to 13.388], Standard Error of Mean 4.830
Statistical Analysis 24: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 7, analysis 21]; Test type: Superiority; p = 0.3741, ANCOVA; LSM Difference = 4.395, 95% CI 2-sided [-5.305 to 14.096], Standard Error of Mean 4.942

8. Secondary Outcome: Change From Baseline in Participant Global Assessment (PGA) of Arthritis at Weeks 1, 2, 4, 8 12 and 16
Description: Participants responded to the question "Considering all the ways your arthritis affects you, how are you feeling today?" was recorded using a 0-100 mm VAS where 0 mm (very well) and 100 mm (very poor). Higher scores indicated worse condition.
Time Frame: Baseline, Week 1, 2, 4, 8, 12 and 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Millimeter (mm)
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
Millimeter (mm)
  Week 1: number analyzed (Participants) | 66 | 71 | 43 | 39 | 72
  Week 1 | -8.160 (2.911) | -19.61 (2.777) | -16.70 (3.633) | -12.53 (3.782) | -5.164 (2.812)
  Week 2: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 2 | -13.66 (2.875) | -18.02 (2.743) | -20.32 (3.608) | -14.99 (3.753) | -9.667 (2.788)
  Week 4: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 4 | -13.21 (2.875) | -20.47 (2.743) | -19.53 (3.608) | -12.74 (3.753) | -10.24 (2.787)
  Week 8: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 8 | -9.062 (2.875) | -21.86 (2.743) | -18.79 (3.608) | -18.09 (3.753) | -12.84 (2.786)
  Week 12: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 12 | -15.54 (2.875) | -21.77 (2.743) | -20.02 (3.608) | -18.54 (3.753) | -11.50 (2.784)
  Week 16: number analyzed (Participants) | 60 | 70 | 38 | 35 | 68
  Week 16 | -13.91 (3.004) | -21.82 (2.789) | -13.29 (3.776) | -13.26 (3.911) | -19.84 (2.854)
Statistical Analysis 1: Comparison: PH-797804, 0.5 mg vs Placebo; Week 1: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 1 as an interaction term, baseline Patient's Global Assessment of Arthritis count as the covariate and participant as a random effect; Test type: Superiority; p = 0.4493, ANCOVA; LSM Difference = -2.996, 95% CI 2-sided [-10.77 to 4.773], Standard Error of Mean 3.958
Statistical Analysis 2: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0002, ANCOVA; LSM Difference = -14.45, 95% CI 2-sided [-22.08 to -6.807], Standard Error of Mean 3.891
Statistical Analysis 3: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0109, ANCOVA; LSM Difference = -11.54, 95% CI 2-sided [-20.42 to -2.661], Standard Error of Mean 4.522
Statistical Analysis 4: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.1137, ANCOVA; LSM Difference = -7.364, 95% CI 2-sided [-16.49 to 1.765], Standard Error of Mean 4.651
Statistical Analysis 5: Comparison: PH-797804, 0.5 mg vs Placebo; Week 2: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 2 as an interaction term, baseline Patient's Global Assessment of Arthritis count as the covariate and participant as a random effect; Test type: Superiority; p = 0.3086, ANCOVA; LSM Difference = -3.989, 95% CI 2-sided [-11.68 to 3.697], Standard Error of Mean 3.915
Statistical Analysis 6: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0303, ANCOVA; LSM Difference = -8.357, 95% CI 2-sided [-15.92 to -0.799], Standard Error of Mean 3.850
Statistical Analysis 7: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0178, ANCOVA; LSM Difference = -10.66, 95% CI 2-sided [-19.47 to -1.845], Standard Error of Mean 4.489
Statistical Analysis 8: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.2486, ANCOVA; LSM Difference = -5.325, 95% CI 2-sided [-14.38 to 3.729], Standard Error of Mean 4.612
Statistical Analysis 9: Comparison: PH-797804, 0.5 mg vs Placebo; Week 4: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 4 as an interaction term, baseline Patient's Global Assessment of Arthritis count as the covariate and participant as a random effect; Test type: Superiority; p = 0.4491, ANCOVA; LSM Difference = -2.965, 95% CI 2-sided [-10.65 to 4.720], Standard Error of Mean 3.915
Statistical Analysis 10: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 8, analysis 9]; Test type: Superiority; p = 0.0081, ANCOVA; LSM Difference = -10.23, 95% CI 2-sided [-17.79 to -2.671], Standard Error of Mean 3.850
Statistical Analysis 11: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 8, analysis 9]; Test type: Superiority; p = 0.0388, ANCOVA; LSM Difference = -9.291, 95% CI 2-sided [-18.10 to -0.480], Standard Error of Mean 4.488
Statistical Analysis 12: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 8, analysis 9]; Test type: Superiority; p = 0.5880, ANCOVA; LSM Difference = -2.500, 95% CI 2-sided [-11.55 to 6.553], Standard Error of Mean 4.611
Statistical Analysis 13: Comparison: PH-797804, 0.5 mg vs Placebo; Week 8: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 8 as an interaction term, baseline Patient's Global Assessment of Arthritis count as the covariate and participant as a random effect; Test type: Superiority; p = 0.3345, ANCOVA; LSM Difference = 3.780, 95% CI 2-sided [-3.904 to 11.464], Standard Error of Mean 3.914
Statistical Analysis 14: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 8, analysis 13]; Test type: Superiority; p = 0.0194, ANCOVA; LSM Difference = -9.019, 95% CI 2-sided [-16.58 to -1.463], Standard Error of Mean 3.849
Statistical Analysis 15: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 8, analysis 13]; Test type: Superiority; p = 0.1855, ANCOVA; LSM Difference = -5.946, 95% CI 2-sided [-14.76 to 2.863], Standard Error of Mean 4.488
Statistical Analysis 16: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 8, analysis 13]; Test type: Superiority; p = 0.2553, ANCOVA; LSM Difference = -5.249, 95% CI 2-sided [-14.30 to 3.803], Standard Error of Mean 4.611
Statistical Analysis 17: Comparison: PH-797804, 0.5 mg vs Placebo; Week 12: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 12 as an interaction term, baseline Patient's Global Assessment of Arthritis count as the covariate and participant as a random effect; Test type: Superiority; p = 0.3020, ANCOVA; LSM Difference = -4.041, 95% CI 2-sided [-11.72 to 3.639], Standard Error of Mean 3.912
Statistical Analysis 18: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 8, analysis 17]; Test type: Superiority; p = 0.0078, ANCOVA; LSM Difference = -10.27, 95% CI 2-sided [-17.82 to -2.715], Standard Error of Mean 3.847
Statistical Analysis 19: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 8, analysis 17]; Test type: Superiority; p = 0.0578, ANCOVA; LSM Difference = -8.522, 95% CI 2-sided [-17.33 to 0.284], Standard Error of Mean 4.486
Statistical Analysis 20: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 8, analysis 17]; Test type: Superiority; p = 0.1270, ANCOVA; LSM Difference = -7.042, 95% CI 2-sided [-16.09 to 2.007], Standard Error of Mean 4.610
Statistical Analysis 21: Comparison: PH-797804, 0.5 mg vs Placebo; Week 16: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 16 as an interaction term, baseline Patient's Global Assessment of Arthritis count as the covariate and participant as a random effect; Test type: Superiority; p = 0.1438, ANCOVA; LSM Difference = 5.927, 95% CI 2-sided [-2.023 to 13.877], Standard Error of Mean 4.051
Statistical Analysis 22: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 8, analysis 21]; Test type: Superiority; p = 0.6149, ANCOVA; LSM Difference = -1.979, 95% CI 2-sided [-9.696 to 5.738], Standard Error of Mean 3.931
Statistical Analysis 23: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 8, analysis 21]; Test type: Superiority; p = 0.1609, ANCOVA; LSM Difference = 6.545, 95% CI 2-sided [-2.610 to 15.700], Standard Error of Mean 4.664
Statistical Analysis 24: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 8, analysis 21]; Test type: Superiority; p = 0.1691, ANCOVA; LSM Difference = 6.579, 95% CI 2-sided [-2.804 to 15.961], Standard Error of Mean 4.780

9. Secondary Outcome: Change From Baseline in Physician Global Assessment of Arthritis at Weeks 1, 2, 4, 8, 12 and 16
Description: Physician assessed the overall impact of arthritis on the participants' daily life based on the disease signs, functional capacity and physical examination. The physician's response was recorded using a 100 mm VAS between 0 mm (very good) and 100 mm (very poor). Higher scores indicating worse condition of arthritis.
Time Frame: Baseline, Week 1, 2, 4, 8, 12 and 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Millimeter (mm)
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
Millimeter (mm)
  Week 1: number analyzed (Participants) | 67 | 71 | 43 | 39 | 72
  Week 1 | -6.612 (2.451) | -10.83 (2.343) | -14.92 (3.053) | -8.898 (3.183) | -5.203 (2.364)
  Week 2: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 2 | -15.87 (2.430) | -17.79 (2.324) | -20.43 (3.032) | -16.15 (3.159) | -10.68 (2.343)
  Week 4: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 4 | -13.91 (2.430) | -20.41 (2.324) | -22.40 (3.032) | -16.23 (3.159) | -13.51 (2.343)
  Week 8: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 8 | -14.44 (2.430) | -24.15 (2.324) | -22.59 (3.032) | -21.38 (3.159) | -13.05 (2.342)
  Week 12: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 12 | -16.90 (2.430) | -23.05 (2.324) | -22.61 (3.032) | -18.80 (3.159) | -13.27 (2.339)
  Week 16: number analyzed (Participants) | 59 | 70 | 38 | 35 | 67
  Week 16 | -19.97 (2.555) | -18.44 (2.364) | -19.21 (3.173) | -18.56 (3.291) | -19.85 (2.409)
Statistical Analysis 1: Comparison: PH-797804, 0.5 mg vs Placebo; Week 1: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 1 as an interaction term, baseline Physician's Global Assessment of Arthritis count as the covariate and participant as a random effect; Test type: Superiority; p = 0.6733, ANCOVA; LSM Difference = -1.409, 95% CI 2-sided [-7.967 to 5.149], Standard Error of Mean 3.341
Statistical Analysis 2: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0859, ANCOVA; LSM Difference = -5.629, 95% CI 2-sided [-12.05 to 0.797], Standard Error of Mean 3.274
Statistical Analysis 3: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0107, ANCOVA; LSM Difference = -9.718, 95% CI 2-sided [-17.18 to -2.259], Standard Error of Mean 3.800
Statistical Analysis 4: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.3463, ANCOVA; LSM Difference = -3.695, 95% CI 2-sided [-11.39 to 4.002], Standard Error of Mean 3.921
Statistical Analysis 5: Comparison: PH-797804, 0.5 mg vs Placebo; Week 2: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 2 as an interaction term, baseline Physician's Global Assessment of Arthritis count as the covariate and participant as a random effect; Test type: Superiority; p = 0.1178, ANCOVA; LSM Difference = -5.185, 95% CI 2-sided [-11.69 to 1.316], Standard Error of Mean 3.312
Statistical Analysis 6: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 9, analysis 5]; Test type: Superiority; p = 0.0288, ANCOVA; LSM Difference = -7.107, 95% CI 2-sided [-13.48 to -0.737], Standard Error of Mean 3.245
Statistical Analysis 7: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 9, analysis 5]; Test type: Superiority; p = 0.0100, ANCOVA; LSM Difference = -9.743, 95% CI 2-sided [-17.15 to -2.340], Standard Error of Mean 3.772
Statistical Analysis 8: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 9, analysis 5]; Test type: Superiority; p = 0.1600, ANCOVA; LSM Difference = -5.468, 95% CI 2-sided [-13.10 to 2.164], Standard Error of Mean 3.888
Statistical Analysis 9: Comparison: PH-797804, 0.5 mg vs Placebo; Week 4: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 4 as an interaction term, baseline Physician's Global Assessment of Arthritis count as the covariate and participant as a random effect; Test type: Superiority; p = 0.9040, ANCOVA; LSM Difference = -0.400, 95% CI 2-sided [-6.900 to 6.101], Standard Error of Mean 3.312
Statistical Analysis 10: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 9, analysis 9]; Test type: Superiority; p = 0.0339, ANCOVA; LSM Difference = -6.895, 95% CI 2-sided [-13.26 to -0.524], Standard Error of Mean 3.245
Statistical Analysis 11: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 9, analysis 9]; Test type: Superiority; p = 0.0186, ANCOVA; LSM Difference = -8.891, 95% CI 2-sided [-16.29 to -1.488], Standard Error of Mean 3.771
Statistical Analysis 12: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 9, analysis 9]; Test type: Superiority; p = 0.4854, ANCOVA; LSM Difference = -2.714, 95% CI 2-sided [-10.35 to 4.918], Standard Error of Mean 3.888
Statistical Analysis 13: Comparison: PH-797804, 0.5 mg vs Placebo; Week 8: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 8 as an interaction term, baseline Physician's Global Assessment of Arthritis count as the covariate and participant as a random effect; Test type: Superiority; p = 0.6753, ANCOVA; LSM Difference = -1.387, 95% CI 2-sided [-7.886 to 5.112], Standard Error of Mean 3.311
Statistical Analysis 14: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 9, analysis 13]; Test type: Superiority; p = 0.0007, ANCOVA; LSM Difference = -11.09, 95% CI 2-sided [-17.46 to -4.724], Standard Error of Mean 3.244
Statistical Analysis 15: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 9, analysis 13]; Test type: Superiority; p = 0.0116, ANCOVA; LSM Difference = -9.535, 95% CI 2-sided [-16.94 to -2.134], Standard Error of Mean 3.771
Statistical Analysis 16: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 9, analysis 13]; Test type: Superiority; p = 0.0326, ANCOVA; LSM Difference = -8.322, 95% CI 2-sided [-15.95 to -0.691], Standard Error of Mean 3.888
Statistical Analysis 17: Comparison: PH-797804, 0.5 mg vs Placebo; Week 12: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 12 as an interaction term, baseline Physician's Global Assessment of Arthritis count as the covariate and participant as a random effect; Test type: Superiority; p = 0.2738, ANCOVA; LSM Difference = -3.624, 95% CI 2-sided [-10.12 to 2.872], Standard Error of Mean 3.309
Statistical Analysis 18: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 9, analysis 17]; Test type: Superiority; p = 0.0026, ANCOVA; LSM Difference = -9.778, 95% CI 2-sided [-16.14 to -3.412], Standard Error of Mean 3.243
Statistical Analysis 19: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 9, analysis 17]; Test type: Superiority; p = 0.0134, ANCOVA; LSM Difference = -9.339, 95% CI 2-sided [-16.74 to -1.941], Standard Error of Mean 3.769
Statistical Analysis 20: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 9, analysis 17]; Test type: Superiority; p = 0.1553, ANCOVA; LSM Difference = -5.528, 95% CI 2-sided [-13.16 to 2.101], Standard Error of Mean 3.886
Statistical Analysis 21: Comparison: PH-797804, 0.5 mg vs Placebo; Week 16: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 16 as an interaction term, baseline Physician's Global Assessment of Arthritis count as the covariate and participant as a random effect; Test type: Superiority; p = 0.9726, ANCOVA; LSM Difference = -0.118, 95% CI 2-sided [-6.878 to 6.641], Standard Error of Mean 3.444
Statistical Analysis 22: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 9, analysis 21]; Test type: Superiority; p = 0.6714, ANCOVA; LSM Difference = 1.409, 95% CI 2-sided [-5.109 to 7.928], Standard Error of Mean 3.321
Statistical Analysis 23: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 9, analysis 21]; Test type: Superiority; p = 0.8693, ANCOVA; LSM Difference = 0.646, 95% CI 2-sided [-7.058 to 8.351], Standard Error of Mean 3.925
Statistical Analysis 24: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 9, analysis 21]; Test type: Superiority; p = 0.7495, ANCOVA; LSM Difference = 1.289, 95% CI 2-sided [-6.631 to 9.208], Standard Error of Mean 4.035

10. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) at Weeks 1, 2, 4, 8, 12 and 16
Description: C-reactive protein is a biochemical measure of inflammation and disease activity.
Time Frame: Baseline, Week 1, 2, 4, 8, 12 and 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: milligram per liter (mg/L)
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
milligram per liter (mg/L)
  Week 1: number analyzed (Participants) | 65 | 70 | 42 | 36 | 69
  Week 1 | -4.785 (3.285) | -10.92 (3.094) | -12.87 (3.953) | -12.06 (4.244) | 4.198 (3.124)
  Week 2: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 2 | -1.077 (3.226) | -6.582 (3.024) | -9.926 (3.880) | -6.835 (4.077) | 2.764 (3.038)
  Week 4: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 4 | 3.492 (3.226) | 0.324 (3.024) | -3.642 (3.880) | 4.182 (4.077) | 2.688 (3.038)
  Week 8: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 8 | 7.190 (3.226) | 3.804 (3.024) | -1.249 (3.880) | 6.727 (4.077) | 3.899 (3.038)
  Week 12: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 12 | 5.468 (3.226) | 0.104 (3.024) | 2.970 (3.880) | 11.585 (4.077) | 2.361 (3.038)
  Week 16: number analyzed (Participants) | 60 | 70 | 38 | 35 | 63
  Week 16 | 1.060 (3.426) | -1.844 (3.093) | -5.559 (4.109) | -4.313 (4.301) | -7.201 (3.234)
Statistical Analysis 1: Comparison: PH-797804, 0.5 mg vs Placebo; Week 1: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 1 as an interaction term, baseline C-Reactive Protein as the covariate and participant as a random effect; Test type: Superiority; p = 0.0447, ANCOVA; LSM Difference = -8.983, 95% CI 2-sided [-17.75 to -0.214], Standard Error of Mean 4.469
Statistical Analysis 2: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.0005, ANCOVA; LSM Difference = -15.12, 95% CI 2-sided [-23.65 to -6.596], Standard Error of Mean 4.345
Statistical Analysis 3: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.0006, ANCOVA; LSM Difference = -17.07, 95% CI 2-sided [-26.84 to -7.296], Standard Error of Mean 4.981
Statistical Analysis 4: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.0019, ANCOVA; LSM Difference = -16.26, 95% CI 2-sided [-26.49 to -6.018], Standard Error of Mean 5.218
Statistical Analysis 5: Comparison: PH-797804, 0.5 mg vs Placebo; Week 2: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 2 as an interaction term, baseline C-Reactive Protein as the covariate and participant as a random effect; Test type: Superiority; p = 0.3792, ANCOVA; LSM Difference = -3.841, 95% CI 2-sided [-12.41 to 4.726], Standard Error of Mean 4.366
Statistical Analysis 6: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p = 0.0276, ANCOVA; LSM Difference = -9.345, 95% CI 2-sided [-17.66 to -1.031], Standard Error of Mean 4.237
Statistical Analysis 7: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p = 0.0093, ANCOVA; LSM Difference = -12.69, 95% CI 2-sided [-22.25 to -3.128], Standard Error of Mean 4.873
Statistical Analysis 8: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p = 0.0566, ANCOVA; LSM Difference = -9.599, 95% CI 2-sided [-19.47 to 0.271], Standard Error of Mean 5.030
Statistical Analysis 9: Comparison: PH-797804, 0.5 mg vs Placebo; Week 4: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 4 as an interaction term, baseline C-Reactive Protein as the covariate and participant as a random effect; Test type: Superiority; p = 0.8540, ANCOVA; LSM Difference = 0.803, 95% CI 2-sided [-7.764 to 9.370], Standard Error of Mean 4.366
Statistical Analysis 10: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 10, analysis 9]; Test type: Superiority; p = 0.5770, ANCOVA; LSM Difference = -2.364, 95% CI 2-sided [-10.68 to 5.950], Standard Error of Mean 4.237
Statistical Analysis 11: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 10, analysis 9]; Test type: Superiority; p = 0.1942, ANCOVA; LSM Difference = -6.330, 95% CI 2-sided [-15.89 to 3.232], Standard Error of Mean 4.873
Statistical Analysis 12: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 10, analysis 9]; Test type: Superiority; p = 0.7665, ANCOVA; LSM Difference = 1.494, 95% CI 2-sided [-8.376 to 11.364], Standard Error of Mean 5.030
Statistical Analysis 13: Comparison: PH-797804, 0.5 mg vs Placebo; Week 8: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 8 as an interaction term, baseline C-Reactive Protein as the covariate and participant as a random effect; Test type: Superiority; p = 0.4512, ANCOVA; LSM Difference = 3.291, 95% CI 2-sided [-5.276 to 11.858], Standard Error of Mean 4.366
Statistical Analysis 14: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 10, analysis 13]; Test type: Superiority; p = 0.9822, ANCOVA; LSM Difference = -0.095, 95% CI 2-sided [-8.409 to 8.220], Standard Error of Mean 4.237
Statistical Analysis 15: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 10, analysis 13]; Test type: Superiority; p = 0.2910, ANCOVA; LSM Difference = -5.148, 95% CI 2-sided [-14.71 to 4.414], Standard Error of Mean 4.873
Statistical Analysis 16: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 10, analysis 13]; Test type: Superiority; p = 0.5741, ANCOVA; LSM Difference = 2.828, 95% CI 2-sided [-7.042 to 12.698], Standard Error of Mean 5.030
Statistical Analysis 17: Comparison: PH-797804, 0.5 mg vs Placebo; Week 12: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 12 as an interaction term, baseline C-Reactive Protein as the covariate and participant as a random effect; Test type: Superiority; p = 0.4768, ANCOVA; LSM Difference = 3.107, 95% CI 2-sided [-5.460 to 11.674], Standard Error of Mean 4.366
Statistical Analysis 18: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 10, analysis 17]; Test type: Superiority; p = 0.5945, ANCOVA; LSM Difference = -2.256, 95% CI 2-sided [-10.57 to 6.058], Standard Error of Mean 4.237
Statistical Analysis 19: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 10, analysis 17]; Test type: Superiority; p = 0.9006, ANCOVA; LSM Difference = 0.609, 95% CI 2-sided [-8.953 to 10.171], Standard Error of Mean 4.873
Statistical Analysis 20: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 10, analysis 17]; Test type: Superiority; p = 0.0670, ANCOVA; LSM Difference = 9.224, 95% CI 2-sided [-0.646 to 19.094], Standard Error of Mean 5.030
Statistical Analysis 21: Comparison: PH-797804, 0.5 mg vs Placebo; Week 16: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 16 as an interaction term, baseline C-Reactive Protein as the covariate and participant as a random effect; Test type: Superiority; p = 0.0757, ANCOVA; LSM Difference = 8.261, 95% CI 2-sided [-0.857 to 17.379], Standard Error of Mean 4.647
Statistical Analysis 22: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 10, analysis 21]; Test type: Superiority; p = 0.2265, ANCOVA; LSM Difference = 5.357, 95% CI 2-sided [-3.329 to 14.043], Standard Error of Mean 4.427
Statistical Analysis 23: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 10, analysis 21]; Test type: Superiority; p = 0.7512, ANCOVA; LSM Difference = 1.642, 95% CI 2-sided [-8.517 to 11.801], Standard Error of Mean 5.178
Statistical Analysis 24: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 10, analysis 21]; Test type: Superiority; p = 0.5876, ANCOVA; LSM Difference = 2.888, 95% CI 2-sided [-7.557 to 13.332], Standard Error of Mean 5.323

11. Secondary Outcome: Change From Baseline in Disease Activity Score in 28 Joints Using 4 Variables (DAS28-4 [CRP]) at Weeks 1, 2, 4, 8, 12 and 16
Description: DAS28-4 (CRP) was calculated from 28-tender joint count and 28-swollen joint count, C-reactive protein (mg/L) and PGA : participant assessed overall disease activity on VAS, score:0(no arthritis) to 100(extreme arthritis). DAS28-4 (CRP) lower than (<) 3.2 implied mild disease activity, 3.2 to 5.1 implied moderate disease activity and greater than (>) 5.1 severe disease activity. Total score range: 0 to 9.4, higher score indicated more disease activity.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12 and 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- PH-797804 ,3 mg: Participants received PH-797804, 3 mg capsule, orally, once daily for 12 weeks. Participants were followed up to 28 days after last dose of study drug. Individual participant participated in the study for a duration of up to 16 weeks.
Arm/Group | PH-797804, 0.5 mg | PH-797804 ,3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
units on a scale
  Week 1: number analyzed (Participants) | 64 | 70 | 42 | 36 | 69
  Week 1 | -0.505 (0.139) | -0.837 (0.131) | -0.928 (0.169) | -0.791 (0.178) | -0.237 (0.132)
  Week 2: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 2 | -0.743 (0.137) | -0.892 (0.129) | -1.101 (0.167) | -0.881 (0.173) | -0.433 (0.130)
  Week 4: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 4 | -0.787 (0.137) | -0.920 (0.129) | -1.062 (0.167) | -0.782 (0.173) | -0.516 (0.130)
  Week 8: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 8 | -0.730 (0.137) | -1.097 (0.129) | -1.077 (0.167) | -0.847 (0.173) | -0.632 (0.130)
  Week 12: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 12 | -1.012 (0.137) | -1.108 (0.129) | -1.174 (0.167) | -0.804 (0.173) | -0.659 (0.130)
  Week 16: number analyzed (Participants) | 62 | 70 | 38 | 36 | 69
  Week 16 | -0.824 (0.145) | -1.013 (0.131) | -0.998 (0.176) | -0.941 (0.181) | -1.095 (0.136)
Statistical Analysis 1: Comparison: PH-797804, 0.5 mg vs Placebo; Week 1: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 1 as an interaction term, baseline DAS28-4(CRP) as the covariate; and participant as a random effect; Test type: Superiority; p = 0.1540, ANCOVA; LSM Difference = -0.269, 95% CI 2-sided [-0.638 to 0.101], Standard Error of Mean 0.188
Statistical Analysis 2: Comparison: PH-797804 ,3 mg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0011, ANCOVA; LSM Difference = -0.600, 95% CI 2-sided [-0.958 to -0.242], Standard Error of Mean 0.182
Statistical Analysis 3: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0011, ANCOVA; LSM Difference = -0.691, 95% CI 2-sided [-1.105 to -0.277], Standard Error of Mean 0.211
Statistical Analysis 4: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0115, ANCOVA; LSM Difference = -0.554, 95% CI 2-sided [-0.983 to -0.125], Standard Error of Mean 0.219
Statistical Analysis 5: Comparison: PH-797804, 0.5 mg vs Placebo; Week 2: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 2 as an interaction term, baseline DAS28-4(CRP) as the covariate; and participant as a random effect; Test type: Superiority; p = 0.0940, ANCOVA; LSM Difference = -0.310, 95% CI 2-sided [-0.673 to 0.053], Standard Error of Mean 0.185
Statistical Analysis 6: Comparison: PH-797804 ,3 mg vs Placebo; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.0109, ANCOVA; LSM Difference = -0.459, 95% CI 2-sided [-0.811 to -0.106], Standard Error of Mean 0.180
Statistical Analysis 7: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.0014, ANCOVA; LSM Difference = -0.667, 95% CI 2-sided [-1.075 to -0.259], Standard Error of Mean 0.208
Statistical Analysis 8: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.0364, ANCOVA; LSM Difference = -0.447, 95% CI 2-sided [-0.867 to -0.028], Standard Error of Mean 0.213
Statistical Analysis 9: Comparison: PH-797804, 0.5 mg vs Placebo; Week 4: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 4 as an interaction term, baseline DAS28-4(CRP) as the covariate; and participant as a random effect; Test type: Superiority; p = 0.1436, ANCOVA; LSM Difference = -0.271, 95% CI 2-sided [-0.634 to 0.092], Standard Error of Mean 0.185
Statistical Analysis 10: Comparison: PH-797804 ,3 mg vs Placebo; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p = 0.0246, ANCOVA; LSM Difference = -0.404, 95% CI 2-sided [-0.757 to -0.052], Standard Error of Mean 0.180
Statistical Analysis 11: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p = 0.0088, ANCOVA; LSM Difference = -0.546, 95% CI 2-sided [-0.954 to -0.138], Standard Error of Mean 0.208
Statistical Analysis 12: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p = 0.2121, ANCOVA; LSM Difference = -0.267, 95% CI 2-sided [-0.686 to 0.152], Standard Error of Mean 0.213
Statistical Analysis 13: Comparison: PH-797804, 0.5 mg vs Placebo; Week 8: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 8 as an interaction term, baseline DAS28-4(CRP) as the covariate; and participant as a random effect; Test type: Superiority; p = 0.5975, ANCOVA; LSM Difference = -0.098, 95% CI 2-sided [-0.461 to 0.265], Standard Error of Mean 0.185
Statistical Analysis 14: Comparison: PH-797804 ,3 mg vs Placebo; [analysis description as in outcome 11, analysis 13]; Test type: Superiority; p = 0.0099, ANCOVA; LSM Difference = -0.464, 95% CI 2-sided [-0.817 to -0.112], Standard Error of Mean 0.180
Statistical Analysis 15: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 11, analysis 13]; Test type: Superiority; p = 0.0328, ANCOVA; LSM Difference = -0.445, 95% CI 2-sided [-0.853 to -0.037], Standard Error of Mean 0.208
Statistical Analysis 16: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 11, analysis 13]; Test type: Superiority; p = 0.3162, ANCOVA; LSM Difference = -0.214, 95% CI 2-sided [-0.633 to 0.205], Standard Error of Mean 0.213
Statistical Analysis 17: Comparison: PH-797804, 0.5 mg vs Placebo; Week 12: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 12 as an interaction term, baseline DAS28-4(CRP) as the covariate; and participant as a random effect; Test type: Superiority; p = 0.0569, ANCOVA; LSM Difference = -0.353, 95% CI 2-sided [-0.716 to 0.010], Standard Error of Mean 0.185
Statistical Analysis 18: Comparison: PH-797804 ,3 mg vs Placebo; [analysis description as in outcome 11, analysis 17]; Test type: Superiority; p = 0.0126, ANCOVA; LSM Difference = -0.449, 95% CI 2-sided [-0.801 to -0.096], Standard Error of Mean 0.180
Statistical Analysis 19: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 11, analysis 17]; Test type: Superiority; p = 0.0135, ANCOVA; LSM Difference = -0.515, 95% CI 2-sided [-0.923 to -0.107], Standard Error of Mean 0.208
Statistical Analysis 20: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 11, analysis 17]; Test type: Superiority; p = 0.4979, ANCOVA; LSM Difference = -0.145, 95% CI 2-sided [-0.564 to 0.274], Standard Error of Mean 0.213
Statistical Analysis 21: Comparison: PH-797804, 0.5 mg vs Placebo; Week 16: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 16 as an interaction term, baseline DAS28-4(CRP) as the covariate; and participant as a random effect; Test type: Superiority; p = 0.1643, ANCOVA; LSM Difference = 0.271, 95% CI 2-sided [-0.111 to 0.653], Standard Error of Mean 0.195
Statistical Analysis 22: Comparison: PH-797804 ,3 mg vs Placebo; [analysis description as in outcome 11, analysis 21]; Test type: Superiority; p = 0.6611, ANCOVA; LSM Difference = 0.081, 95% CI 2-sided [-0.282 to 0.445], Standard Error of Mean 0.185
Statistical Analysis 23: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 11, analysis 21]; Test type: Superiority; p = 0.6587, ANCOVA; LSM Difference = 0.097, 95% CI 2-sided [-0.333 to 0.526], Standard Error of Mean 0.219
Statistical Analysis 24: Comparison: PH-797804, 0.5 mg vs Placebo; [analysis description as in outcome 11, analysis 21]; Test type: Superiority; p = 0.4903, ANCOVA; LSM Difference = 0.154, 95% CI 2-sided [-0.284 to 0.592], Standard Error of Mean 0.223

12. Secondary Outcome: Number of Participants Who Withdrew From Study Due to Lack of Efficacy
Time Frame: Baseline up to Week 16
Population: FAS included all participants randomized to treatment and who had taken at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
Participants | 9 | 3 | 3 | 2 | 6

13. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Weeks 1, 2, 4, 8, 12 and 16
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dressing/grooming, arising, eating, walking, reaching, gripping, hygiene, and "other common activities" over past week. Each item scored on 4-point scale from 0 to 3: 0= no difficulty; 1= some difficulty; 2= much difficulty; 3= unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total average possible score range 0 (least difficulty) to 3 (extreme difficulty), where higher scores indicate more difficulty while performing daily living activities.
Time Frame: Baseline, Week 1, 2, 4, 8, 12 and 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
units on a scale
  Week 1: number analyzed (Participants) | 66 | 71 | 43 | 39 | 72
  Week 1 | -0.166 (0.066) | -0.323 (0.064) | -0.291 (0.083) | -0.144 (0.086) | -0.046 (0.064)
  Week 2: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 2 | -0.286 (0.065) | -0.341 (0.063) | -0.370 (0.082) | -0.201 (0.086) | -0.151 (0.063)
  Week 4: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 4 | -0.241 (0.065) | -0.343 (0.063) | -0.405 (0.082) | -0.258 (0.086) | -0.186 (0.063)
  Week 8: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 8 | -0.159 (0.065) | -0.409 (0.063) | -0.391 (0.082) | -0.192 (0.086) | -0.219 (0.063)
  Week 12: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Week 12 | -0.253 (0.065) | -0.433 (0.063) | -0.356 (0.082) | -0.142 (0.086) | -0.220 (0.063)
  Week 16: number analyzed (Participants) | 60 | 70 | 38 | 37 | 69
  Week 16 | -0.263 (0.068) | -0.280 (0.064) | -0.245 (0.086) | -0.210 (0.089) | -0.346 (0.065)
Statistical Analysis 1: Comparison: PH-797804, 0.5 mg vs Placebo; Week 1: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 1 as an interaction term, baseline HAQ-DI as the covariate and participant as a random effect; Test type: Superiority; p = 0.1857, ANCOVA; LSM Difference = -0.119, 95% CI 2-sided [-0.296 to 0.057], Standard Error of Mean 0.090
Statistical Analysis 2: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0019, ANCOVA; LSM Difference = -0.277, 95% CI 2-sided [-0.451 to -0.103], Standard Error of Mean 0.089
Statistical Analysis 3: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0178, ANCOVA; LSM Difference = -0.244, 95% CI 2-sided [-0.446 to -0.042], Standard Error of Mean 0.103
Statistical Analysis 4: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.3547, ANCOVA; LSM Difference = -0.098, 95% CI 2-sided [-0.305 to 0.110], Standard Error of Mean 0.106
Statistical Analysis 5: Comparison: PH-797804, 0.5 mg vs Placebo; Week 2: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 2 as an interaction term, baseline HAQ-DI as the covariate and participant as a random effect; Test type: Superiority; p = 0.1301, ANCOVA; LSM Difference = -0.135, 95% CI 2-sided [-0.310 to 0.040], Standard Error of Mean 0.089
Statistical Analysis 6: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 13, analysis 5]; Test type: Superiority; p = 0.0313, ANCOVA; LSM Difference = -0.190, 95% CI 2-sided [-0.363 to -0.017], Standard Error of Mean 0.088
Statistical Analysis 7: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 13, analysis 5]; Test type: Superiority; p = 0.0323, ANCOVA; LSM Difference = -0.219, 95% CI 2-sided [-0.420 to -0.019], Standard Error of Mean 0.102
Statistical Analysis 8: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 13, analysis 5]; Test type: Superiority; p = 0.6318, ANCOVA; LSM Difference = -0.050, 95% CI 2-sided [-0.256 to 0.156], Standard Error of Mean 0.105
Statistical Analysis 9: Comparison: PH-797804, 0.5 mg vs Placebo; Week 4: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 4 as an interaction term, baseline HAQ-DI as the covariate and participant as a random effect; Test type: Superiority; p = 0.5388, ANCOVA; LSM Difference = -0.055, 95% CI 2-sided [-0.230 to 0.120], Standard Error of Mean 0.089
Statistical Analysis 10: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 13, analysis 9]; Test type: Superiority; p = 0.0755, ANCOVA; LSM Difference = -0.157, 95% CI 2-sided [-0.329 to 0.016], Standard Error of Mean 0.088
Statistical Analysis 11: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 13, analysis 9]; Test type: Superiority; p = 0.0323, ANCOVA; LSM Difference = -0.219, 95% CI 2-sided [-0.420 to -0.019], Standard Error of Mean 0.102
Statistical Analysis 12: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 13, analysis 9]; Test type: Superiority; p = 0.4948, ANCOVA; LSM Difference = -0.072, 95% CI 2-sided [-0.277 to 0.134], Standard Error of Mean 0.105
Statistical Analysis 13: Comparison: PH-797804, 0.5 mg vs Placebo; Week 8: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 8 as an interaction term, baseline HAQ-DI as the covariate and participant as a random effect; Test type: Superiority; p = 0.5022, ANCOVA; LSM Difference = 0.060, 95% CI 2-sided [-0.115 to 0.235], Standard Error of Mean 0.089
Statistical Analysis 14: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 13, analysis 13]; Test type: Superiority; p = 0.0307, ANCOVA; LSM Difference = -0.190, 95% CI 2-sided [-0.363 to -0.018], Standard Error of Mean 0.088
Statistical Analysis 15: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 13, analysis 13]; Test type: Superiority; p = 0.0933, ANCOVA; LSM Difference = -0.172, 95% CI 2-sided [-0.372 to 0.029], Standard Error of Mean 0.102
Statistical Analysis 16: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 13, analysis 13]; Test type: Superiority; p = 0.7967, ANCOVA; LSM Difference = 0.027, 95% CI 2-sided [-0.179 to 0.233], Standard Error of Mean 0.105
Statistical Analysis 17: Comparison: PH-797804, 0.5 mg vs Placebo; Week 12: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 12 as an interaction term, baseline HAQ-DI as the covariate and participant as a random effect; Test type: Superiority; p = 0.7059, ANCOVA; LSM Difference = -0.034, 95% CI 2-sided [-0.208 to 0.141], Standard Error of Mean 0.089
Statistical Analysis 18: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 13, analysis 17]; Test type: Superiority; p = 0.0154, ANCOVA; LSM Difference = -0.213, 95% CI 2-sided [-0.386 to -0.041], Standard Error of Mean 0.088
Statistical Analysis 19: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 13, analysis 17]; Test type: Superiority; p = 0.1836, ANCOVA; LSM Difference = -0.136, 95% CI 2-sided [-0.336 to 0.065], Standard Error of Mean 0.102
Statistical Analysis 20: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 13, analysis 17]; Test type: Superiority; p = 0.4577, ANCOVA; LSM Difference = 0.078, 95% CI 2-sided [-0.128 to 0.284], Standard Error of Mean 0.105
Statistical Analysis 21: Comparison: PH-797804, 0.5 mg vs Placebo; Week 16: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 16 as an interaction term, baseline HAQ-DI as the covariate and participant as a random effect; Test type: Superiority; p = 0.3692, ANCOVA; LSM Difference = 0.082, 95% CI 2-sided [-0.098 to 0.262], Standard Error of Mean 0.092
Statistical Analysis 22: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 13, analysis 21]; Test type: Superiority; p = 0.4677, ANCOVA; LSM Difference = 0.065, 95% CI 2-sided [-0.111 to 0.241], Standard Error of Mean 0.090
Statistical Analysis 23: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 13, analysis 21]; Test type: Superiority; p = 0.3427, ANCOVA; LSM Difference = 0.100, 95% CI 2-sided [-0.107 to 0.307], Standard Error of Mean 0.106
Statistical Analysis 24: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 13, analysis 21]; Test type: Superiority; p = 0.2120, ANCOVA; LSM Difference = 0.135, 95% CI 2-sided [-0.077 to 0.347], Standard Error of Mean 0.108

14. Secondary Outcome: Change From Baseline in Modified Brief Pain Inventory-Short Form (mBPI-SF) Score at Weeks 1, 2, 4, 8 and 12
Description: The modified brief pain inventory-short form (mBPI-SF) is a pain assessment tool used to measure both pain intensity and pain interference using an 11-point numeric rating scale. Participants rated their pain severity, using a scale from 0 (no pain) to 10 (pain as bad as you can imagine), where higher scores indicate greater intensity of pain. Participants also rated the level of pain interference using a scale from 0 (no interference) to 10 (complete interference), where higher scores indicate more degree of interference in general daily activities.
Time Frame: Baseline, Week 1, 2, 4, 8 and 12
Population: FAS included all participants randomized to treatment and who had taken at least 1 dose of study medication. Here, 'number analyzed' signifies participants evaluable for this outcome measure at specified time points. Missing values were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
units on a scale
  Pain Intensity: Week 1: number analyzed (Participants) | 66 | 71 | 43 | 39 | 71
  Pain Intensity: Week 1 | -0.671 (0.247) | -1.140 (0.236) | -1.190 (0.309) | -0.926 (0.325) | -0.083 (0.239)
  Pain Intensity: Week 2: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Pain Intensity: Week 2 | -0.929 (0.244) | -1.069 (0.233) | -1.507 (0.307) | -1.004 (0.323) | -0.487 (0.237)
  Pain Intensity: Week 4: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Pain Intensity: Week 4 | -0.788 (0.244) | -1.360 (0.233) | -1.489 (0.307) | -1.069 (0.323) | -0.640 (0.237)
  Pain Intensity: Week 8: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Pain Intensity: Week 8 | -0.640 (0.244) | -1.383 (0.233) | -1.379 (0.307) | -0.870 (0.323) | -0.616 (0.237)
  Pain Intensity: Week 12: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Pain Intensity: Week 12 | -0.937 (0.244) | -1.556 (0.233) | -0.983 (0.307) | -1.024 (0.323) | -0.460 (0.237)
  Pain Interference:Week 1: number analyzed (Participants) | 66 | 71 | 43 | 39 | 71
  Pain Interference:Week 1 | -0.889 (0.265) | -1.266 (0.253) | -1.290 (0.331) | -1.057 (0.349) | -0.376 (0.257)
  Pain Interference:Week 2: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Pain Interference:Week 2 | -1.275 (0.262) | -1.306 (0.251) | -1.752 (0.329) | -1.227 (0.347) | -0.735 (0.255)
  Pain Interference:Week 4: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Pain Interference:Week 4 | -1.181 (0.262) | -1.426 (0.251) | -1.782 (0.329) | -1.150 (0.347) | -0.961 (0.255)
  Pain Interference:Week 8: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Pain Interference:Week 8 | -0.736 (0.262) | -1.574 (0.251) | -1.702 (0.329) | -1.187 (0.347) | -0.754 (0.255)
  Pain Interference:Week 12: number analyzed (Participants) | 69 | 74 | 44 | 40 | 74
  Pain Interference:Week 12 | -1.030 (0.262) | -1.615 (0.251) | -1.433 (0.329) | -1.187 (0.347) | -0.820 (0.255)
Statistical Analysis 1: Comparison: PH-797804, 0.5 mg vs Placebo; Week 1: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 1 as an interaction term, baseline Pain Intensity Domain of mBPI as the covariate; and participant as a random effect; Test type: Superiority; p = 0.0815, ANCOVA; LSM Difference = -0.587, 95% CI 2-sided [-1.248 to 0.074], Standard Error of Mean 0.337
Statistical Analysis 2: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.0015, ANCOVA; LSM Difference = -1.057, 95% CI 2-sided [-1.707 to -0.407], Standard Error of Mean 0.331
Statistical Analysis 3: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.0042, ANCOVA; LSM Difference = -1.107, 95% CI 2-sided [-1.863 to -0.351], Standard Error of Mean 0.385
Statistical Analysis 4: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.0348, ANCOVA; LSM Difference = -0.842, 95% CI 2-sided [-1.624 to -0.060], Standard Error of Mean 0.398
Statistical Analysis 5: Comparison: PH-797804, 0.5 mg vs Placebo; Week 2: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 2 as an interaction term, baseline Pain Intensity Domain of mBPI as the covariate; and participant as a random effect; Test type: Superiority; p = 0.1843, ANCOVA; LSM Difference = -0.442, 95% CI 2-sided [-1.095 to 0.211], Standard Error of Mean 0.332
Statistical Analysis 6: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 14, analysis 5]; Test type: Superiority; p = 0.0760, ANCOVA; LSM Difference = -0.582, 95% CI 2-sided [-1.225 to 0.061], Standard Error of Mean 0.327
Statistical Analysis 7: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 14, analysis 5]; Test type: Superiority; p = 0.0078, ANCOVA; LSM Difference = -1.019, 95% CI 2-sided [-1.769 to -0.270], Standard Error of Mean 0.382
Statistical Analysis 8: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 14, analysis 5]; Test type: Superiority; p = 0.1905, ANCOVA; LSM Difference = -0.517, 95% CI 2-sided [-1.292 to 0.258], Standard Error of Mean 0.395
Statistical Analysis 9: Comparison: PH-797804, 0.5 mg vs Placebo; Week 4: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 4 as an interaction term, baseline Pain Intensity Domain of mBPI as the covariate; and participant as a random effect; Test type: Superiority; p = 0.6552, ANCOVA; LSM Difference = -0.149, 95% CI 2-sided [-0.801 to 0.504], Standard Error of Mean 0.332
Statistical Analysis 10: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 14, analysis 9]; Test type: Superiority; p = 0.0281, ANCOVA; LSM Difference = -0.720, 95% CI 2-sided [-1.363 to -0.078], Standard Error of Mean 0.327
Statistical Analysis 11: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 14, analysis 9]; Test type: Superiority; p = 0.0263, ANCOVA; LSM Difference = -0.850, 95% CI 2-sided [-1.599 to -0.100], Standard Error of Mean 0.382
Statistical Analysis 12: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 14, analysis 9]; Test type: Superiority; p = 0.2772, ANCOVA; LSM Difference = -0.429, 95% CI 2-sided [-1.204 to 0.346], Standard Error of Mean 0.395
Statistical Analysis 13: Comparison: PH-797804, 0.5 mg vs Placebo; Week 8: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 8 as an interaction term, baseline Pain Intensity Domain of mBPI as the covariate; and participant as a random effect; Test type: Superiority; p = 0.9433, ANCOVA; LSM Difference = -0.024, 95% CI 2-sided [-0.676 to 0.629], Standard Error of Mean 0.332
Statistical Analysis 14: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 14, analysis 13]; Test type: Superiority; p = 0.193, ANCOVA; LSM Difference = -0.768, 95% CI 2-sided [-1.410 to -0.125], Standard Error of Mean 0.327
Statistical Analysis 15: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 14, analysis 13]; Test type: Superiority; p = 0.461, ANCOVA; LSM Difference = -0.763, 95% CI 2-sided [-1.512 to -0.013], Standard Error of Mean 0.382
Statistical Analysis 16: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 14, analysis 13]; Test type: Superiority; p = 0.5200, ANCOVA; LSM Difference = -0.254, 95% CI 2-sided [-1.029 to 0.521], Standard Error of Mean 0.395
Statistical Analysis 17: Comparison: PH-797804, 0.5 mg vs Placebo; Week 12: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 12 as an interaction term, baseline Pain Intensity Domain of mBPI as the covariate; and participant as a random effect; Test type: Superiority; p = 0.1526, ANCOVA; LSM Difference = -0.476, 95% CI 2-sided [-1.129 to 0.177], Standard Error of Mean 0.332
Statistical Analysis 18: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 14, analysis 17]; Test type: Superiority; p = 0.0009, ANCOVA; LSM Difference = -1.095, 95% CI 2-sided [-1.738 to -0.453], Standard Error of Mean 0.327
Statistical Analysis 19: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 14, analysis 17]; Test type: Superiority; p = 0.1711, ANCOVA; LSM Difference = -0.523, 95% CI 2-sided [-1.273 to 0.227], Standard Error of Mean 0.382
Statistical Analysis 20: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 14, analysis 17]; Test type: Superiority; p = 0.1539, ANCOVA; LSM Difference = -0.563, 95% CI 2-sided [-1.338 to 0.211], Standard Error of Mean 0.395
Statistical Analysis 21: Comparison: PH-797804, 0.5 mg vs Placebo; Week 1: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 1 as an interaction term, baseline Pain Interference Domain of mBPI as the covariate; and participant as a random effect; Test type: Superiority; p = 0.1554, ANCOVA; LSM Difference = -0.512, 95% CI 2-sided [-1.219 to 0.195], Standard Error of Mean 0.360
Statistical Analysis 22: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 14, analysis 21]; Test type: Superiority; p = 0.0124, ANCOVA; LSM Difference = -0.889, 95% CI 2-sided [-1.585 to -0.193], Standard Error of Mean 0.354
Statistical Analysis 23: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 14, analysis 21]; Test type: Superiority; p = 0.0268, ANCOVA; LSM Difference = -0.914, 95% CI 2-sided [-1.723 to -0.106], Standard Error of Mean 0.412
Statistical Analysis 24: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 14, analysis 21]; Test type: Superiority; p = 0.1113, ANCOVA; LSM Difference = -0.681, 95% CI 2-sided [-1.519 to 0.158], Standard Error of Mean 0.427
Statistical Analysis 25: Comparison: PH-797804, 0.5 mg vs Placebo; Week 2: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 2 as an interaction term, baseline Pain Interference Domain of mBPI as the covariate; and participant as a random effect; Test type: Superiority; p = 0.1305, ANCOVA; LSM Difference = -0.540, 95% CI 2-sided [-1.240 to 0.160], Standard Error of Mean 0.356
Statistical Analysis 26: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 14, analysis 25]; Test type: Superiority; p = 0.1043, ANCOVA; LSM Difference = -0.571, 95% CI 2-sided [-1.261 to 0.118], Standard Error of Mean 0.351
Statistical Analysis 27: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 14, analysis 25]; Test type: Superiority; p = 0.0131, ANCOVA; LSM Difference = -1.017, 95% CI 2-sided [-1.820 to -0.214], Standard Error of Mean 0.409
Statistical Analysis 28: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 14, analysis 25]; Test type: Superiority; p = 0.2459, ANCOVA; LSM Difference = -0.492, 95% CI 2-sided [-1.324 to 0.340], Standard Error of Mean 0.424
Statistical Analysis 29: Comparison: PH-797804, 0.5 mg vs Placebo; Week 4: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 4 as an interaction term, baseline Pain Interference Domain of mBPI as the covariate; and participant as a random effect; Test type: Superiority; p = 0.5360, ANCOVA; LSM Difference = -0.221, 95% CI 2-sided [-0.921 to 0.479], Standard Error of Mean 0.356
Statistical Analysis 30: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 14, analysis 29]; Test type: Superiority; p = 0.1858, ANCOVA; LSM Difference = -0.465, 95% CI 2-sided [-1.155 to 0.225], Standard Error of Mean 0.351
Statistical Analysis 31: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 14, analysis 29]; Test type: Superiority; p = 0.0451, ANCOVA; LSM Difference = -0.821, 95% CI 2-sided [-1.624 to -0.018], Standard Error of Mean 0.409
Statistical Analysis 32: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 14, analysis 29]; Test type: Superiority; p = 0.6551, ANCOVA; LSM Difference = -0.189, 95% CI 2-sided [-1.021 to 0.643], Standard Error of Mean 0.424
Statistical Analysis 33: Comparison: PH-797804, 0.5 mg vs Placebo; Week 8: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 8 as an interaction term, baseline Pain Interference Domain of mBPI as the covariate; and participant as a random effect; Test type: Superiority; p = 0.9602, ANCOVA; LSM Difference = 0.018, 95% CI 2-sided [-0.682 to 0.718], Standard Error of Mean 0.356
Statistical Analysis 34: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 14, analysis 33]; Test type: Superiority; p = 0.0198, ANCOVA; LSM Difference = -0.820, 95% CI 2-sided [-1.510 to -0.131], Standard Error of Mean 0.351
Statistical Analysis 35: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 14, analysis 33]; Test type: Superiority; p = 0.0208, ANCOVA; LSM Difference = -0.948, 95% CI 2-sided [-1.751 to -0.145], Standard Error of Mean 0.409
Statistical Analysis 36: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 14, analysis 33]; Test type: Superiority; p = 0.3077, ANCOVA; LSM Difference = -0.433, 95% CI 2-sided [-1.265 to 0.400], Standard Error of Mean 0.424
Statistical Analysis 37: Comparison: PH-797804, 0.5 mg vs Placebo; Week 12: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 12 as an interaction term, baseline Pain Interference Domain of mBPI as the covariate; and participant as a random effect; Test type: Superiority; p = 0.5550, ANCOVA; LSM Difference = -0.211, 95% CI 2-sided [-0.911 to 0.490], Standard Error of Mean 0.356
Statistical Analysis 38: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 14, analysis 37]; Test type: Superiority; p = 0.0239, ANCOVA; LSM Difference = -0.795, 95% CI 2-sided [-1.485 to -0.106], Standard Error of Mean 0.351
Statistical Analysis 39: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 14, analysis 37]; Test type: Superiority; p = 0.1342, ANCOVA; LSM Difference = -0.613, 95% CI 2-sided [-1.416 to 0.190], Standard Error of Mean 0.409
Statistical Analysis 40: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 14, analysis 37]; Test type: Superiority; p = 0.3868, ANCOVA; LSM Difference = -0.367, 95% CI 2-sided [-1.199 to 0.465], Standard Error of Mean 0.424

15. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Version 2 at Weeks 4 and 12
Description: The SF-36 version 2 is a 36-item generic health status measure standardized survey is a standardized survey evaluating 8 domains of functional health and well-being: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE) and mental health (MH). The summary score of these concepts is summarized as Physical component summary (PCS) score and Mental component summary (MCS) score, are based on a normalized sum of the 8 scale scores PF, RP, BP, GH, VT, SF, RE, and MH. The score for each of 8 domains were scaled from 0 (lowest level of functioning) to100 (highest level of functioning, where higher scores represented better level of functioning. 8 domains were summarized as 2 summary scores; PCS and MCS. Score range for each of the 2 summary scores = 0 (lowest level of functioning) to 100 (highest level of functioning), where higher scores represented better level of functioning.
Time Frame: Baseline, Weeks 4, 12
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
units on a scale
  Week 4: PCS: number analyzed (Participants) | 68 | 72 | 41 | 37 | 72
  Week 4: PCS | 2.374 (0.806) | 3.509 (0.777) | 5.778 (1.051) | 2.818 (1.074) | 1.582 (0.785)
  Week 12: PCS: number analyzed (Participants) | 68 | 73 | 41 | 39 | 73
  Week 12: PCS | 2.857 (0.806) | 4.277 (0.773) | 4.525 (1.051) | 2.031 (1.056) | 1.763 (0.781)
  Week 4: MCS: number analyzed (Participants) | 68 | 72 | 41 | 37 | 72
  Week 4: MCS | 1.676 (1.198) | 3.870 (1.144) | 4.897 (1.570) | 3.408 (1.602) | 2.579 (1.167)
  Week 12: MCS: number analyzed (Participants) | 68 | 73 | 41 | 39 | 73
  Week 12: MCS | 0.556 (1.198) | 2.656 (1.137) | 2.761 (1.570) | 2.341 (1.572) | 0.131 (1.161)
Statistical Analysis 1: Comparison: PH-797804, 0.5 mg vs Placebo; Week 4: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 4 as an interaction term, baseline SF-36 PCS as the covariate; and participant as a random effect; Test type: Superiority; p = 0.4693, ANCOVA; LSM Difference = 0.792, 95% CI 2-sided [-1.357 to 2.941], Standard Error of Mean 1.093
Statistical Analysis 2: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.0743, ANCOVA; LSM Difference = 1.927, 95% CI 2-sided [-0.190 to 4.044], Standard Error of Mean 1.077
Statistical Analysis 3: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.0012, ANCOVA; LSM Difference = 4.196, 95% CI 2-sided [1.668 to 6.723], Standard Error of Mean 1.286
Statistical Analysis 4: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.3452, ANCOVA; LSM Difference = 1.236, 95% CI 2-sided [-1.335 to 3.807], Standard Error of Mean 1.308
Statistical Analysis 5: Comparison: PH-797804, 0.5 mg vs Placebo; Week 12: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 12 as an interaction term, baseline SF-36 PCS as the covariate; and participant as a random effect; Test type: Superiority; p = 0.3162, ANCOVA; LSM Difference = 1.095, 95% CI 2-sided [-1.050 to 3.239], Standard Error of Mean 1.091
Statistical Analysis 6: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 15, analysis 5]; Test type: Superiority; p = 0.0195, ANCOVA; LSM Difference = 2.514, 95% CI 2-sided [0.406 to 4.622], Standard Error of Mean 1.072
Statistical Analysis 7: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 15, analysis 5]; Test type: Superiority; p = 0.0320, ANCOVA; LSM Difference = 2.762, 95% CI 2-sided [0.239 to 5.285], Standard Error of Mean 1.283
Statistical Analysis 8: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 15, analysis 5]; Test type: Superiority; p = 0.8356, ANCOVA; LSM Difference = 0.268, 95% CI 2-sided [-2.268 to 2.804], Standard Error of Mean 1.290
Statistical Analysis 9: Comparison: PH-797804, 0.5 mg vs Placebo; Week 4: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 4 as an interaction term, baseline SF-36 MCS as the covariate; and participant as a random effect; Test type: Superiority; p = 0.5787, ANCOVA; LSM Difference = -0.904, 95% CI 2-sided [-4.101 to 2.293], Standard Error of Mean 1.626
Statistical Analysis 10: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 15, analysis 9]; Test type: Superiority; p = 0.4203, ANCOVA; LSM Difference = 1.291, 95% CI 2-sided [-1.854 to 4.436], Standard Error of Mean 1.600
Statistical Analysis 11: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 15, analysis 9]; Test type: Superiority; p = 0.2272, ANCOVA; LSM Difference = 2.318, 95% CI 2-sided [-1.449 to 6.084], Standard Error of Mean 1.916
Statistical Analysis 12: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 15, analysis 9]; Test type: Superiority; p = 0.6707, ANCOVA; LSM Difference = 0.829, 95% CI 2-sided [-2.998 to 4.655], Standard Error of Mean 1.947
Statistical Analysis 13: Comparison: PH-797804, 0.5 mg vs Placebo; Week 12: Estimates and p-values based on repeated measures analysis of covariance with treatment, country and week as fixed effects, treatment Week 12 as an interaction term, baseline SF-36 MCS as the covariate; and participant as a random effect; Test type: Superiority; p = 0.7935, ANCOVA; LSM Difference = 0.425, 95% CI 2-sided [-2.764 to 3.613], Standard Error of Mean 1.622
Statistical Analysis 14: Comparison: PH-797804, 3 mg vs Placebo; [analysis description as in outcome 15, analysis 13]; Test type: Superiority; p = 0.1135, ANCOVA; LSM Difference = 2.525, 95% CI 2-sided [-0.605 to 5.655], Standard Error of Mean 1.592
Statistical Analysis 15: Comparison: PH-797804, 6 mg vs Placebo; [analysis description as in outcome 15, analysis 13]; Test type: Superiority; p = 0.1697, ANCOVA; LSM Difference = 2.630, 95% CI 2-sided [-1.128 to 6.388], Standard Error of Mean 1.912
Statistical Analysis 16: Comparison: PH-797804, 10 mg vs Placebo; [analysis description as in outcome 15, analysis 13]; Test type: Superiority; p = 0.2500, ANCOVA; LSM Difference = 2.210, 95% CI 2-sided [-1.561 to 5.981], Standard Error of Mean 1.918

16. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent events are events between first dose of study drug and up to week 16 after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious AEs.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all participants randomized to treatment who had taken at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
Participants
  AEs | 38 | 47 | 31 | 33 | 42
  SAEs | 2 | 3 | 4 | 5 | 1

17. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Haemoglobin, haematocrit, red blood cell count less than(<) 0.8*lower limit of normal [LLN], platelets <0.5*LLN and (&) greater than(>) 1.75*ULN, white blood cell count <0.6*LLN&>1.5x ULN, lymphocytes <0.8*LLN&>1.2*ULN, total neutrophils <0.8*LLN&>1.2*ULN, basophils, eosinophils, monocytes >1.2*ULN; total bilirubin >1.5*ULN, aspartate aminotransferase, alanine aminotransferase, gamma glutamyl transferase, alkaline phosphatase >3.0*ULN, total protein <0.8*LLN&>1.2*ULN, albumin <0.8*LLN&>1.2*ULN; blood urea nitrogen, Creatinine, Uric Acid >1.2*ULN; Cholesterol >1.3*ULN, HDL Cholesterol <0.8*LLN, LDL Cholesterol >1.2*ULN, Triglycerides >1.3*ULN; Electrolytes: sodium <0.95*LLN&>1.05*ULN, potassium <0.9*LLN&>1.1*ULN, chloride, calcium, magnesium, bicarbonate <0.9*LLN&>1.1*ULN, phosphate <0.8*LLN&>1.2x ULN; glucose <0.6*LLN&>1.5*ULN, human chorionic gonadotrophin >0; CRP >1.25*ULN, ([urine-RBC, WBC, epithelial cells, crystals, yeast cells] >=6), urine casts >1, urine Bacteria >20.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all participants randomized to treatment who had taken at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
Participants | 68 | 72 | 43 | 40 | 74

18. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Pre-defined criteria for vital sign abnormalities: Maximum (max) increase from baseline in supine systolic blood pressure (SBP) >=30 milliliters of mercury (mmHg), maximum increase from baseline in supine diastolic blood pressure (DBP) >=20 mmHg.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all participants randomized to treatment who had taken at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
Participants
  Max Increase from Baseline in Supine SBP | 4 | 6 | 4 | 7 | 8
  Max Increase from Baseline in Supine DBP | 4 | 9 | 2 | 8 | 9

19. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in 12-Lead Electrocardiogram (ECG) Parameters
Description: 12-lead ECG were performed after the participant had rested quietly for at least 10 minutes in a supine position. ECG parameters included RR interval, PR interval, QRS complex, QT interval, corrected QT (QTc) interval, Bazett's correction QT (QTcB) interval, Heart Rate and Fridericia's correction (QTcF) interval. Clinical significance of 12-Lead ECG was judged by investigator.
Time Frame: Baseline up to Week 16
Population: FAS included all participants randomized to treatment and who had taken at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
Participants | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Criteria for ECG abnormalities: maximum QT interval (millisecond [msec]): < 450, 450 to <480, 480 to <500, >= 500; maximum QT interval with Bazett's correction (QTcB interval) (msec): <450, 450 to <480, 480 to <500, >=500; maximum QT interval with Fridericia's correction (QTcF interval) (msec): <450, 450 to <480, 480 to <500, >=500; maximum QTc interval increase from baseline (msec): change <30, 30 <=change <60, change >=60.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all participants randomized to treatment who had taken at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
Participants
  Maximum QT Interval (<450 msec) | 65 | 58 | 39 | 32 | 68
  Maximum QT Interval (450 to <480 msec) | 4 | 11 | 5 | 6 | 7
  Maximum QT Interval (480 to <500 msec) | 0 | 4 | 0 | 0 | 0
  Maximum QT Interval (>=500 msec) | 0 | 1 | 0 | 2 | 0
  Maximum QTcB Interval (<450 msec) | 54 | 46 | 32 | 25 | 61
  Maximum QTcB Interval (450 to <480 msec) | 14 | 24 | 12 | 15 | 13
  Maximum QTcB Interval (480 to <500 msec) | 1 | 3 | 0 | 0 | 1
  Maximum QTcB Interval (>=500 msec) | 0 | 1 | 0 | 0 | 0
  Maximum QTcF Interval (<450 msec) | 66 | 58 | 40 | 30 | 73
  Maximum QTcF Interval (450 to <480 msec) | 3 | 14 | 4 | 10 | 2
  Maximum QTcF Interval (480 to <500 msec) | 0 | 2 | 0 | 0 | 0
  Maximum QTcF Interval (>=500 msec) | 0 | 0 | 0 | 0 | 0
  QTc Interval increase from baseline(change < 30 msec) | 57 | 62 | 36 | 34 | 70
  QTc Interval increase from baseline(change 30 msec to <60 msec) | 11 | 11 | 8 | 6 | 5
  QTc Interval increase from baseline(change >=60 msec) | 1 | 1 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Clinically Significant Physical Examination Abnormalities
Description: Following criteria and body systems were examined to identify the clinically significant physical examination abnormalities; general appearance, skin (presence of rash), head, ears, eyes, nose, and throat, lungs (auscultation), heart (auscultation for presence of murmurs, gallops, rubs, peripheral edema), abdominal (palpation and auscultation), neurologic (mental status, station, gait, reflexes, motor and sensory function, coordination). Physical examination abnormalities were as determined by the investigator.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all participants randomized to treatment who had taken at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
Participants | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Minimum Observed Plasma Pre-dose Concentration (Ctrough Min) of Steady State
Time Frame: Predose
Population: Analysis set included all participants randomized to treatment who had taken at least 1 dose of PH-797804.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Groups:
- PH-797804, 3 mg: Participants received PH-797804, 3 mg capsule, orally, once daily for 12 weeks. Participants were followed up to 28 days after last dose of study drug Individual participant participated in the study for a duration of up to 16 weeks.
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg
Number analyzed (Participants) | 69 | 74 | 44 | 40
Nanogram per milliliter | 5.4 (1.8) | 30.8 (8.9) | 51.3 (15.9) | 79.4 (26.4)

23. Secondary Outcome: Number of Participants With Concomitant Medications
Description: Concomitant medication (any medication other than, and in addition to, the study medication) taken for any period of time during the study and was coded by World Health Organization (WHO) medical dictionary.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all participants randomized to treatment who had taken at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PH-797804, 0.5 mg | PH-797804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Number analyzed (Participants) | 69 | 74 | 44 | 40 | 75
Participants | 69 | 73 | 44 | 40 | 74

ADVERSE EVENTS:
Time Frame: Baseline up to Week 16
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as nonserious in another participant or 1 participant may have experienced both serious and nonserious event during study. Safety population.
Arm/Group | PH-797804, 0.5 mg | PH79804, 3 mg | PH-797804, 6 mg | PH-797804, 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/69 | 3/74 | 4/44 | 5/40 | 1/75
Other Adverse Events (participants affected / at risk) | 38/69 | 45/74 | 27/44 | 32/40 | 41/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PH-797804, 0.5 mg (N=69) | PH79804, 3 mg (N=74) | PH-797804, 6 mg (N=44) | PH-797804, 10 mg (N=40) | Placebo (N=75)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0
Cyclitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Electrocardiogram change (Investigations) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PH-797804, 0.5 mg (N=69) | PH79804, 3 mg (N=74) | PH-797804, 6 mg (N=44) | PH-797804, 10 mg (N=40) | Placebo (N=75)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 2 | 2 | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 4 | 7 | 4
Nausea (Gastrointestinal disorders) | 2 | 3 | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 3 | 1 | 0 | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 3
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 4 | 0 | 2 | 0
Flatulance (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 4 | 1 | 0 | 0 | 2
Mass (General disorders) | 1 | 0 | 0 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 2 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Neurosis (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 4 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 3 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0 | 3
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 1 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 2 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 5 | 1 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Chloasma (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Palpable purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1 | 1 | 5 | 2
Gastroenteritis (Infections and infestations) | 2 | 2 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 4 | 2 | 2 | 2
Parotitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 3 | 0 | 3 | 5
Paronychia (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 3 | 7 | 1 | 2 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1
Tinea versicolour (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 3 | 0 | 1 | 2
Cystitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Vulvovaginitis (Infections and infestations) | 0 | 1 | 1 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 2 | 0 | 0 | 1 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 2 | 2 | 1 | 5 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 2 | 2 | 0 | 2
Cervical root pain (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 1 | 1 | 0
Radiculitis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Allergic pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 3 | 4 | 2
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Accelerated hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 1 | 1 | 0
Episcleritis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0
Corneal erosion (Eye disorders) | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fractured ischium (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 2
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 1 | 2
Electrocardiogram Q wave abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 2
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urethritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 2 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.